# The GlaxoSmithKline group of companies

| Division | : Worldwide Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for 200812: A phase IIIB, 24-week randomised, double-blind study to compare 'closed' triple therapy (FF/UMEC/VI) with 'open' triple therapy (FF/VI + UMEC), in subjects with chronic obstructive pulmonary disease (COPD) |
|---|---|---|
| Compound Number | : | GSK2834425 (GW685698, GSK573719, GW642444) |
| <b>Effective Date</b> | : | 22-JUN-2017 |

# **Author's Name and Functional Area:**

| PPD | |
|--------------------------------------------------------------|-------------|
| Principal Statistician, Statistics and Programming (Clinical | 13-Jun-2017 |
| Statistics) | |
| PPD | 13-Jun-2017 |
| Manager, Statistics | |

# Approved by:

| PPD | | 22-JUN-2017 |
|--------------|------------------------------------------------|-------------|
| Director, St | atistics and Programming (Clinical Statistics) | 22-JUN-201/ |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited

# **TABLE OF CONTENTS**

| | | | | ŀ | PAGE |
|---|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS | S PLAN SYNPOSIS | 5 |
| 2. | SUMN | MARY OF | KEY PRO | TOCOL INFORMATION | 7 |
| | 2.1. | | | otocol Defined Statistical Analysis Plan | |
| | 2.2. | | | and Endpoint(s) | |
| | 2.3. | Study D | esigní | | 8 |
| | 2.4. | | | ses | |
| 3. | PLAN | NED ANA | LYSES | | 10 |
| | 3.1. | Final An | alyses | | 10 |
| 4. | ANAL | YSIS POF | PULATION | S | 11 |
| | 4.1. | | | S | |
| 5. | | ENTIONS/<br>Handling | Sg of Missing | DATA ANALYSES AND DATA HANDLING Dataom Additional Subset Populations | 13 |
| 6. | CTUD | V DODLII | ATIONI AN | IALYSES | 4.5 |
| 0. | 6.1. | | | ed Analyses | |
| | 0.1. | 6.1.1. | | on | |
| | | 6.1.2. | | ant Medications | |
| | | 6.1.3. | | t Compliance | |
| | | 6.1.4. | | Characteristics | |
| | | 6.1.5. | | alfunction | |
| 7. | PRIMA | ARY STA | TISTICAL | ANALYSES | 17 |
| | 7.1. | | | | |
| | | 7.1.1. ´ | | of Planned Efficacy Analyses | |
| | | | 7.1.1.1. | Spirometry data | |
| | | 7.1.2. | Planned l | Efficacy Statistical Analyses | |
| 8. | SECO | NDARY S | STATISTIC | AL ANALYSES | 21 |
| | 8.1. | Other Ef | ficacy Ana | lyses | 21 |
| | | 8.1.1. | | of Planned Efficacy Analyses | |
| | | | 8.1.1.1. | St. George's Respiratory Questionnaire for | |
| | | | | COPD Patients (SGRQ-C) | 22 |
| | | | 8.1.1.2. | COPD Exacerbations | 22 |
| | | | 8.1.1.3. | Baseline Dyspnea Index (BDI)/Transitional | |
| | | | | Dyspnea Index (TDI) Focal Score | |
| | | 8.1.2. | | Other Efficacy Statistical Analyses | |
| | | | 8.1.2.1. | SGRQ Total Score | |
| | | | 8.1.2.2. | TDI | 23 |
| | | | 8.1.2.3. | Proportion of Responders according to SGRQ | |
| | | | _ , _ | Total Score and Responders according to TDI | |
| | | | 8.1.2.4. | COPD Exacerbations | |
| | 8.2. | | | | |
| | | 8.2.1. | Overview | of Planned Analyses | 25 |

| | | | | CONFIDENTIAL | |
|---|---|---|---|---|---|
| | | | | 2 | 200812 |
| | | | 8.2.1.1. | Adverse Events of Special Interest | 28 |
| | | | 8.2.1.2. | Pneumonia | |
| | | | 8.2.1.3. | Vital Signs | |
| | | | 8.2.1.4. | ECGs | |
| | | 1 | 8.2.1.5. | Pregnancy | 29 |
| 9. | REFE | RENCES | | | 30 |
| 10 | ADDE | UDICES | | | 21 |
| 10. | 10.1. | | | ol Deviation Management and Definitions for | 31 |
| | | | | | 32 |
| | | 10.1.1. | Exclusion | of Data from the ITT Analyses | 32 |
| | | | | s from mPP Population | |
| | 10.2. | | | Events | |
| | 10.3. | | | ment Windows | |
| | 10.4. | | | ent States and Phases | |
| | | 10.4.1. | Treatment | Phase for Concomitant Medication Data | 38 |
| | | 10.4.2. | Treatment | Phase for Other Data | 39 |
| | 10.5. | Appendix | 5: Data Di | splay Standards & Handling Conventions | 41 |
| | | 10.5.1. | Study Trea | atment & Sub-group Display Descriptors | 41 |
| | | 10.5.2. | Baseline D | Definition & Derivations | 41 |
| | | | 10.5.2.1. | Baseline Definitions | 41 |
| | | 10.5.3. | Reporting | Process & Standards | 42 |
| | 10.6. | | | I and Transformed Data | |
| | | 10.6.1. | General | | 44 |
| | | | | ulation | |
| | | | | nd Health Outcomes | |
| | 10.7. | | | ure Withdrawals & Handling of Missing Data | |
| | | | | Withdrawals | |
| | | | | of Missing Data | |
| | | | | Handling of Missing or Partial Dates | |
| | | | 10.7.2.2. | Handling of Missing Data for Statistical | |
| | | | | Analysis | |
| | 10.8. | | | nter Studies | |
| | | | | or Handling Centers | |
| | 10.9. | | | ation of Covariates, Subgroups & Other Strata | |
| | | | | of Covariates, Subgroups & Other Strata | |
| | 10.10. | Appendix | 10: Multip | le Comparisons & Multiplicity | 60 |

10.10.1. Handling of Multiple Comparisons & Multiplicity.......60

 10.13.1. Data Display Numbering
 64

 10.13.2. Programming Note
 64

 10.13.3. Study Population Tables
 65

 10.13.4. Study Population Figures
 66

 10.13.5. Efficacy Tables
 66

 10.13.6. Efficacy Figures
 67

10.12. Appendix 12: Abbreviations .......62

10.13. Appendix 13: List of Data Displays......64

10.11. Appendix 11: Model Checking and Diagnostics for Statistical

# CONFIDENTIAL

| 10.13.7. | Safety Tables | 68 |
|----------|-------------------|----|
| | Safety Figures | |
| | ICH Listings | |
| | .Non-ICH Listings | |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP details all planned analyses and outputs required for the final Clinical Study Report (CSR) of study 200812 |
| Protocol | This RAP is based on the protocol amendment (Dated: 29-June-2016) of study 200812 (GSK Document Number. 2015N261999_03) and eCRF Version 2.1 |
| Primary<br>Objective | To compare the effect of FF/UMEC/VI with FF/VI + UMEC on lung function after 24 weeks of treatment in COPD subjects |
| Primary | Change from baseline in trough FEV1 at Week 24 |
| Endpoint | The primary treatment comparison of FF/UMEC/VI with FF/VI+UMEC will be performed on trough FEV1 at Week 24, for the mPP Population. |
| Secondary<br>Objectives | <ul> <li>To compare the effects of FF/UMEC/VI with FF/VI + UMEC on health related quality of life and dyspnoea after 24 weeks of treatment</li> <li>To compare the effect of FF/UMEC/VI with FF/VI + UMEC on time to first moderate or severe exacerbation during 24 weeks of treatment</li> </ul> |
| Secondary<br>Endpoints | <ul> <li>Proportion of Responders based on the St George Respiratory Questionnaire (SGRQ) Total Score at Week 24</li> <li>Change from baseline in SGRQ Total Score at Week 24</li> <li>Proportion of Responders based on Transitional Dyspnoea Index (TDI) focal score at Week 24</li> <li>TDI focal score at Week 24</li> <li>Time to first moderate/severe exacerbation</li> </ul> |
| Study<br>Design | <ul> <li>This is a phase IIIB, 24-week, randomised, double-blind, parallel group, multicenter study evaluating FF/UMEC/VI (100/62.5/25mcg) delivered via a single ELLIPTA ('closed' triple) plus matching placebo ELLIPTA versus FF/VI (100/25mcg) + UMEC (62.5mcg) delivered via two ELLIPTAs ('open' triple), all taken once daily.</li> <li>Subjects will be randomized 1:1 to either FF/UMEC/VI or FF/VI+UMEC. The</li> </ul> |
| | randomisation will be stratified based on long-acting bronchodilator usage during the run-in (none, one or two long-acting bronchodilators per day). |
| | <ul> <li>A study with 816 evaluable subjects for the primary analysis will have 90% power to determine non-inferiority of FF/UMEC/VI to FF/VI+UMEC based on trough FEV1 at Week 24, an estimate of residual standard deviation (SD) for trough FEV1 at Week 24 of 220mL, at the one-sided 2.5% significance level when the margin of non-inferiority is 50mL and the true mean treatment difference is assumed to be 0mL.</li> </ul> |
| | Based on approximately 20% of subjects who are randomized discontinuing study treatment or being excluded from the mPP population at Week 24, approximately 1020 subjects will be randomised |
| Planned<br>Analyses | No interim analyses are planned for this study. |

| Overview | Key Elements of the RAP |
|---|---|
| | <ul> <li>All decisions regarding final analysis, as defined in this RAP document, will be<br/>made by Source Data Lock (SDL) prior to Study Data Tabulation Model (SDTM)<br/>Database Freeze (DBF) of the study data except for the identification of<br/>protocol deviation (PD) that require treatment details. The PD of taking<br/>incorrect treatment and treatment non-compliance (based on active treatment)<br/>will be identified following DBF.</li> </ul> |
| Analysis<br>Populations | <ul> <li>All Subjects Enrolled (ASE) population includes all subjects, for whom a record<br/>exists in the study database, including screen failures and any subject who was<br/>not screened but experienced an SAE between the date of informed consent<br/>and the planned date of the Screening visit. All Subjects Enrolled population<br/>(ASE) will be used for subject disposition, reason for withdrawal prior to<br/>randomisation, inclusion, exclusion and randomisation criteria deviations and<br/>SAEs for non randomised subjects.</li> </ul> |
| | <ul> <li>Intent-to-treat (ITT) population, which comprises all randomized subjects,<br/>excluding those who were randomized in error. A subject who is recorded as a<br/>screen or run-in failure and also randomized will be considered to be<br/>randomized in error. Any other subject who receives a randomisation number<br/>will be considered to have been randomized. Intent-to-treat (ITT) population will<br/>be used for study population, efficacy and safety endpoints.</li> </ul> |
| | <ul> <li>Modified Per-Protocol (mPP) population includes all subjects in the ITT<br/>Population who do not have a full protocol deviation considered to impact<br/>efficacy.</li> </ul> |
| | <ul> <li>Data following a moderate or severe COPD exacerbation or pneumonia<br/>will be excluded from analysis due to the potential impact of the<br/>exacerbation or the medications used to treat it</li> </ul> |
| | <ul> <li>Subjects with partial protocol deviations considered to impact efficacy<br/>will be included in the mPP Population but will have their data excluded<br/>from analyses from the time of deviation onwards</li> </ul> |
| | <ul> <li>mPP population will be used for the primary treatment comparison of<br/>the primary endpoint only.</li> </ul> |
| Hypothesis | The null hypothesis is that the difference in trough FEV1 between treatment groups is less than or equal to a pre-specified non-inferiority margin $-\Delta$ : |
| | $H_0$ : T1 $-$ T2 $\leq$ $-\Delta$ |
| | The alternative hypothesis is that the difference between treatment groups is greater than the margin. |
| | H1: T1 – T2 > -Δ |
| | where T1 and T2 are the treatment means for FF/UMEC/VI and FF/VI+UMEC, respectively. |
| | The non-inferiority margin has been set at 50mL, which is half the generally accepted minimal clinically important difference (MCID) for trough FEV1. |
| | If the lower bound of the two-sided 95% confidence interval around the |

| Overview | Key Elements of the RAP |
|---|---|
| | (FF/UMEC/VI vs. FF/VI+UMEC) treatment difference is above -50mL then FF/UMEC/VI will be considered non-inferior to FF/VI+UMEC. |
| Primary<br>Analyses | The primary endpoint of change from baseline in trough FEV1 at Week 24 will be analyzed in the mPP population, using a mixed model repeated measures (MMRM) analysis, including trough FEV1 recorded at each of Week 4, 12 and 24. The model will include covariates of stratum (number of long-acting bronchodilators per day during the run-in, baseline FEV1, Visit, geographical region, treatment and Visit by baseline interaction. A Visit by treatment interaction term will also be included to allow treatment effects to be estimated at each visit separately. The variance-covariance matrix will be assumed unstructured. |
| Other<br>Efficacy<br>Analyses | The MMRM analysis will be repeated for the ITT Population |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There was one change to the originally planned statistical analysis specified in the protocol.

The Adherent population in the originally planned statistical analysis specified in the protocol is now referred to as the Modified Per Protocol (MPP) population. This is simply a change of the name of population. The definition remains the same.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objective | Primary Endpoint |
| To compare the effect of FF/UMEC/VI with FF/VI + UMEC on lung function after 24 weeks of treatment | Change from baseline in trough FEV1 at Week 24 |
| | Other Endpoints |
| | <ul> <li>Change from baseline in trough FEV1 on Week 4 and 12</li> <li>Change from baseline in trough FVC on Week 4,12 and 24</li> </ul> |
| Secondary Objective | Secondary Endpoint |
| To compare the effects of<br>FF/UMEC/VI with FF/VI + UMEC on<br>health related quality of life and<br>dyspnoea after 24 weeks of treatment | <ul> <li>Proportion of Responders based on the St George<br/>Respiratory Questionnaire (SGRQ) Total Score at Week<br/>24</li> <li>Change from baseline in SGRQ Total Score at Week 24</li> <li>Proportion of Responders based on Transitional</li> </ul> |
| To compare the effect of FF/UMEC/VI with FF/VI + UMEC on time to first moderate or severe exacerbation | Dyspnoea Index (TDI) focal score at Week 24 TDI focal score at Week 24 |

| Objectives | Endpoints |
|---|---|
| during 24 weeks of treatment | Time to first moderate or severe exacerbation |
| | Other Endpoints |
| | <ul> <li>Proportion of Responders based on the St George<br/>Respiratory Questionnaire (SGRQ) Total Score at Week<br/>12</li> <li>Change from baseline in SGRQ Total Score at Week 12</li> <li>Proportion of Responders based on TDI focal score at<br/>Week 12</li> <li>TDI focal score at Week 12</li> </ul> |
| PK | |
| To compare the PK of FF, UMEC and<br>VI when given as FF/UMEC/VI or<br>FF/VI+UMEC in a subset of subjects | Population PK (in a subset of approximately 180 subjects) (note: Population PK analysis is subject to a separate RAP) |
| Safety | |
| To compare the safety profile of<br>FF/UMEC/VI with FF/VI + UMEC over<br>24 weeks of treatment | <ul> <li>Incidence of adverse events</li> <li>Incidence of adverse events of special interest</li> <li>ECG measurements</li> <li>Vital signs</li> <li>Haematological and clinical chemistry parameters</li> </ul> |

# 2.3. Study Design



| Overview of Study I | Design and Key Features |
|---|---|
| Design Features | This is a phase IIIB, 24-week, randomised, double-blind, parallel group, multicenter study evaluating FF/UMEC/VI delivered via a single ELLIPTA ('closed' triple) plus matching placebo ELLIPTA versus FF/VI + UMEC delivered via two ELLIPTAs ('open' triple), all taken once daily. |
| | Subjects will be randomized 1:1 to either FF/UMEC/VI or FF/VI+UMEC. The randomisation will be stratified based on long-acting bronchodilator usage during the run-in (none, one or two long-acting bronchodilators per day). |
| | Subjects will run-in on their existing COPD medications for 2 weeks and in addition will be provided with short acting albuterol/salbutamol to be used on an as-needed basis (rescue medication) throughout the study. Subjects will discontinue all existing COPD medications at the start of the randomised treatment period but may continue their study-supplied rescue albuterol/salbutamol. |
| | A subject will be considered to have completed the study when they have completed all phases of the study including screening, run-in, the randomised treatment phase, and safety follow-up. Subjects who stop study treatment early will complete an Early Withdrawal Visit, followed by a Safety Follow-Up a week later and be withdrawn from the study. |
| | <ul> <li>Approximately 180 subjects, in selected sites, will be asked to participate in PK research. There will be two PK groups (subset A and subset B). Approximately 120 subjects will be assigned to subset A and approximately 60 subjects will be assigned to subset B. Subjects in subset A will provide a blood sample at two time-points at Week 12 (V4) and at Week 24 (V5). Subjects in subset B will provide bloodsamples at seven time points at Week 12 (V4).</li> </ul> |
| | <ul> <li>A subset of subjects in selected countries (Russia, Japan and<br/>Germany) providing PK samples for subset A will also be asked to<br/>take part in a hair sample scalp &amp; finger secretion PK Sub-Study.<br/>Hair sample scalp &amp; finger secretion PK data is subject to a<br/>separate RAP.</li> </ul> |
| Dosing | The ELLIPTA contains 30 doses (FF/UMEC/VI, FF/VI, UMEC or placebo) and subjects will be instructed to administer one dose from each ELLIPTA once daily in the morning. |
| Treatment Assignment | <ul> <li>Following the run-in period, subjects who fulfil the randomisation criteria<br/>will be randomised (1:1) to one of the following double-blind treatment<br/>groups for 24 weeks:</li> </ul> |
| | FF/UMEC/VI 100/62.5/25mcg and placebo, both via the ELLIPTA once daily in the morning or, |
| | FF/VI 100/25mcg and UMEC 62.5mcg, both via the ELLIPTA once daily in the morning |

| Overview of Study | Desi | gn and Key Features |
|---|---|---|
| | <ul> <li>GSK RandAll NG used to generate randomisation schedules.</li> </ul> | |
| | • | Country based randomisation for treatment allocation. |
| | • | The randomisation is stratified based on long-acting bronchodilator usage during the run-in (none, one or two long-acting bronchodilators per day). |
| Interim Analysis | • | No interim analysis is planned for the study. |

# 2.4. Statistical Hypotheses

The primary objective of this study is to compare FF/UMEC/VI with FF/VI+UMEC in COPD subjects. The primary endpoint is change from baseline in trough FEV1 at Week 24. The primary analysis is the comparison of this endpoint for FF/UMEC/VI vs. FF/VI+UMEC.

The null hypothesis is that the difference in change from baseline trough FEV1 between treatment groups is less than or equal to a pre-specified non-inferiority margin  $-\Delta$ :

H0: T1 − T2 ≤ 
$$-\Delta$$

The alternative hypothesis is that the difference between treatments is greater than the margin:

$$H_1: T_1 - T_2 > -\Delta$$

where  $T_1$  and  $T_2$  are the treatment means for FF/UMEC/VI and FF/VI+UMEC, respectively.

The non-inferiority margin has been set at 50mL, which is half the generally accepted minimal clinically important difference (MCID) for trough FEV1.

If the lower bound of the two-sided 95% confidence interval around the (FF/UMEC/VI vs. FF/VI+UMEC) treatment difference is above -50mL then FF/UMEC/VI will be considered non-inferior to FF/VI+UMEC.

#### 3. PLANNED ANALYSES

# 3.1. Final Analyses

No interim analysis is planned for this study. The final planned analyses will be performed after the completion of the following sequential steps (for this Clinical Data Interchange Standards Consortium [CDISC] study):

- 1. All subjects have completed the study or been withdrawn as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (SDL) has been declared by Data Management on System Independent (SI) datasets.

- 3. SI data to SDTM data conversion has completed by Conversion Service and quality control of SDTM has completed by DM.
- 4. Study is unblinded by Clinical Statistician in Randall NG.
- 5. Clinical Programmer extracts unblinded randomization and container codes from Randall NG and SMS2000 file from SMS2000 and then unblinds relevant SDTM datasets (Example: DM, EX, SE, PC etc) as per Clinical Statistics & Programming Study and Subject Treatment Unblinding Guideline document.
- 6. Database freeze on SDTM datasets has been declared by DM.

Note: following database frozen (*i.e.*, treatment unblinding), protocol deviations for subject received incorrect treatment and for non-compliance based on active treatment will be identified and flagged as PP exclusionary. These protocol deviations will be flagged as PP exclusionary in ADaM DV dataset.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects | All subjects for whom a record exists in the | Subject Disposition |
| Enrolled (ASE) | study database, including screen failures and any subject who was not screened but experienced an SAE between the date of informed consent and the planned date of the | Reason for withdrawal prior to randomisation |
| | Screening visit. | Inclusion, exclusion<br>and randomisation<br>criteria deviations |
| | | SAEs for non-<br>randomised<br>subjects |
| Intent-to-Treat | All randomized subjects, excluding those who | Study Population |
| (ITT) | were randomized in error. A subject who is recorded as a screen or run-in failure and also | Efficacy |
| | randomized will be considered to be randomized in error. Any other subject who | Health-related Quality of Life |
| | receives a randomization number will be considered to have been randomized. | Inhaler Assessments |
| | | Safety |
| Modified Per<br>Protocol (mPP) | <ul> <li>All subjects in the ITT Population who do not have a full protocol deviation considered to impact efficacy.</li> <li>Data following a moderate/severe COPD exacerbation or pneumonia will be excluded from analysis due to the potential impact of the exacerbation or the medications used to treat it</li> </ul> | Primary treatment<br>comparison of the<br>primary endpoint<br>only |
| | Subjects with partial protocol deviations considered to impact efficacy will be included | |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | in the mPP Population but will have their data excluded from analyses from the time of deviation onwards. | |

**NOTES :** Please refer to Appendix 13: List of Data Displays which details the population to be used for each displays being generated.

In the event one or more investigators are withdrawn from the study due to concerns over protocol deviation then a further population will be defined which will consist of all subjects in the ITT population excluding subjects from those investigative sites. This population will be used to perform additional sensitivity analysis for the primary efficacy endpoint only, and will only be defined if the combined enrolment at these sites exceeds  $\geq 2\%$  of the overall ITT study enrolment.

### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Exclusions from the mPP analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for mPP Population).
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to SDTM DBF to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- Subjects who received an incorrect container will be captured as an important
  protocol deviation. Whether or not the incorrect container contains incorrect
  treatment will be identified following DBF in the Analysis Data Model (ADaM)
  dataset. Overall treatment non-compliance based on active treatment will also be
  identified following DBF and will be flagged as PP exclusionary in ADaM DV
  dataset.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.
- A listing of any treatment misallocations will be produced for the ASE Population.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Treatment States and Phases |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 10.8 | Appendix 8: Multicenter Studies |
| 10.9 | Appendix 9: Examination of Covariates, Subgroups & Other Strata |
| 10.10 | Appendix 10: Multiple Comparisons & Multiplicity |
| 10.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses. |
| 10.12 | Appendix 12: Abbreviations & Trade Marks |
| 10.13 | Appendix 13: List of Data Displays |

# 5.1. Handling of Missing Data

The primary estimand for this study is a 'de jure' estimand. The primary analysis will use an 'MPP' population, using only data collected on-treatment and excluding data following protocol deviation or other event considered to impact the primary efficacy endpoint of change from baseline in trough FEV1 (as detailed in Section 10.1.2). This will evaluate the treatment difference if all subjects had taken the treatment as directed in the protocol which is considered the appropriate estimand for a determination of non-inferiority.

All data excluded from the primary efficacy analysis will be assumed to be missing at random. The sensitivity of the results to this assumption will be investigated by use of a 'tipping point' analysis as described in Section 7.1.2. This will evaluate various assumptions for the mean change from baseline in trough FEV1 for data excluded from the primary analysis, including scenarios where the response to treatment on FF/UMEC/VI is worse than that on FF/VI + UMEC and vice versa.

An alternative estimand will be evaluated. This will use the ITT population using all data collected on-treatment, for the change from baseline in trough FEV1. (No off-treatment

data for trough FEV1 were collected in this study.) All missing data will be assumed to be missing at random. This will evaluate the treatment difference in all randomized subjects, regardless of adherence to the protocol but assuming the treatment effect for subjects who discontinued treatment was similar to that for those who completed treatment.

# 5.2. Handling of Data from Additional Subset Populations

Approximately 180 subjects, in selected sites, will be asked to participate in the PK analysis. There will be two PK groups (subset A and subset B). Approximately 120 subjects will be assigned to subset A and approximately 60 subjects will be assigned to subset B. Subjects in subset A will provide a blood sample at two time-points at Week 12 (V4) and at Week 24 (V5). Subjects in subset B will provide blood samples at seven time points at Week 12 (V4).

Population PK analysis population (including subjects provided blood PK samples from this study and other studies in Closed Triple Program) will be described in a separate RAP.

A subset of subjects in selected countries (Russia, Japan and Germany) providing PK samples for subset A will also be asked to take part in a hair sample scalp & finger secretion PK Sub-Study. Separate analysis populations will be defined for the hair sample scalp & finger PK and analysis will be described in a separate RAP.

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses generally will be based on the ITT population unless otherwise specified. Displays which use the ASE population or mPP population are identified below.

Table 2 provides an overview of the planned study population analyses, with the detailed list of data displays being presented in Section 10.13.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Study Populations and Reasons for Screen/Run-in | <b>Y</b> 1 | | Υ |
| Failures | 1 | | ı |
| Attendance at Clinic Visits | Υ | | |
| Study Treatment Status | Υ | | Y |
| End of Study Record | Y | <b>Y</b> <sup>2</sup> | Y |
| Number of Subjects | <b>Y</b> 3 | | |
| Inclusion and Exclusion Criteria Deviations | <b>Y</b> 4 | | Υ4 |
| Important Protocol Deviations | Υ | | Y |
| Exclusion from Modified Per Protocol Population | Υ | | Y |
| Reasons for study withdrawal | | | Υ |
| Demography | | 1 | 1 |
| Demographic Characteristics | <b>Y</b> 5,7 | | Y |
| Race and Racial Combination | <b>Y</b> 7 | | Υ |
| Medical Conditions | | | 1 |
| Medical Conditions (Current/Past ) | Υ | | Y |
| Cardiovascular Risk Factors | Υ | | |
| Family History of Cardiovascular Risk Factors | Υ | | Y |
| Smoking History at Screening | Υ | | Y |
| Smoking Status | Υ | | Υ |
| Disease Characteristics | | • | L |
| COPD Exacerbation History | Υ | | Υ |
| Screening Lung Function | <b>Y</b> 5,7 | | Υ |
| Reversibility and GOLD Grade(1-4) at Screening | <b>Y</b> 7 | | Υ |
| CAT Score at Screening | Υ | | Υ |
| Concomitant Medications | | | |
| COPD Medications | <b>Y</b> 6 | | Υ |
| COPD Medication Combination at Screening | <b>Y</b> <sup>7</sup> | | |
| Non-COPD Medications | Y8 | | Υ |
| Relationship between ATC Level1/Ingredient/Verbatim | | | Y |
| Text for Non-COPD Medications | | | I |
| Long-acting Bronchodilator Usage Per Day During Run-in (Randomisation Strata) | <b>Y</b> 7,9 | | Y |

| Display Type | Data | Displays Gene | rated |
|---|---|---|---|
| | Table | Figure | Listing |
| Treatment Compliance | | | |
| Treatment Compliance | Υ | | Y |
| Study Population Listings | | | |
| Randomized and Actual Treatments | | | Y |
| Treatment Blind Broken During Study | | | Y |
| Treatment Misallocations | | | Y |
| Randomisation Strata (Derived and from eCRF) | | | Y |
| Percent Oxygen in Blood | | | Y |
| Inhaler Malfunction | | | Y |

#### NOTES:

- Y = Yes display generated.
- 1. ASE population
- 2. Kaplan-Meier plot
- 3. By country (ASE population); by age category (ASE population); by geographical region, country and centre (ITT population)
- 4. Screen failures (ASE population) and ITT population separately
- 5. Repeat by country (ITT population)
- 6. Run-in/On-treatment/Post-treatment and Given for Reasons other than an Exacerbation, given for an exacerbation, separately
- 7. ITT population and mPP population separately
- 8. On-treatment and Post-treatment, separately
- 9. None, one or two long acting bronchodilator

# 6.1.1. Disposition

The study population summary will show the number of subjects overall who were enrolled, the number of pre-screen failures, the number of screen and run-in failures and the number with each reason for screen or run-in failure, the number of subjects in each treatment group and overall who were randomized, in the ITT population and the number of subjects in the mPP population.

The end of study record summary shows the number of subjects who completed the study as well as the number who withdrew early from the study along with reasons for early withdrawal.

The summary of study treatment status shows the number of subjects who completed study treatment as well as the number who stopped study treatment prior to the end of the study, along with the reasons for discontinuation.

#### 6.1.2. Concomitant Medications

COPD concomitant medications that have been stopped prior to Screening and non-COPD concomitant medications that have been stopped prior to randomization will be listed and not be included in any summary tables.

Non-COPD medication tables will report by Anatomical Therapeutic Chemical (ATC) level 1 and ingredient. COPD medication tables will report by respiratory medication class (RMC) and ingredient (See Section 10.6.2).

Multi-ingredient medications will be presented according to their combination ATC classification rather than the classification of the ingredients.

The number and percentage of subjects taking each medication in the RMC categories ICS, LABA, LAMA, PDE4 inhibitors, Xanthines and combinations of these RMCs on the day of the Screening visit will be presented.

The number of long-acting bronchodilator used per day during the run-in (none, one or two long-acting bronchodilators per day) will be summarised.

### 6.1.3. Treatment Compliance

Treatment compliance will be determined as discussed in Section 10.6.2. Note that the ELLIPTA inhaler used to dispense FF/UMEC/VI, FF/VI, UMEC or placebo has a counter that shows exactly the number of doses remaining. Compliance will be calculated based on the count recored on the dose counter and will be calculated overall and separately for each ELLIPTA inhaler (the inhaler contains FF/UMEC/VI or FF/VI and the inhaler contains placebo or UMEC).

#### 6.1.4. Disease Characteristics

The screening lung function summary will include pre-bronchodilator and post-salbutamol FEV1, FVC, FEV1/FVC ratio, FEV1 as a percentage of predicted normal, and FEV1 reversibility to salbutamol (expressed in milliliters [mL] and as a percentage).

#### 6.1.5. Inhaler Malfunction

Device malfunction occurs during the study will be recorded in eCRF with container numbers. This data will be listed.

# 7. PRIMARY STATISTICAL ANALYSES

# 7.1. Efficacy Analyses

## 7.1.1. Overview of Planned Efficacy Analyses

The primary efficacy analyses for change from baseline in Trough FEV1 will be on the mPP population. All outputs produced for the primary endpoint will be repeated on the ITT population.

Table 3 provides an overview of the planned efficacy analyses for Trough FEV1, with full details of data displays being presented in Section 10.13, List of Data Displays.

Other endpoints of trough FEV1 at Weeks 4 and 12, and trough FVC at Weeks 4, 12 and 24 are also included in this section as they are related to the primary endpoint.

Table 3 Overview of Planned Efficacy Analyses

| | | Absolute | | | | | | | | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Analy | sis ( | Sumn | Summary | | Individual | | Stats Analysis | | | Summary | | Individual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Spirometry | | | | | | | | | | | | | | |
| Baseline FEV1 | | | | <b>Y</b> 1 | | | Y <sup>2</sup> | | | | | | | |
| Trough FEV1 | <b>Y</b> 1 | | | <b>Y</b> 1 | | | Y <sup>2</sup> | <b>Y</b> 1 | Y <sup>4</sup> | | <b>Y</b> 1 | <b>Y</b> 4,5 | | Y <sup>2</sup> |
| (MMRM analysis) | | | | | | | | | | | | | | |
| Trough FVC | | | | <b>Y</b> 3 | | | Y <sup>2</sup> | | | | <b>Y</b> 3 | | | Y <sup>2</sup> |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - 1. For mPP population and ITT population, separately.
  - 2. ITT population only and include a flag for mPP population.
  - 3. ITT population only
  - 4. MPP population only
  - 5. empirical distribution function plot

# 7.1.1.1. Spirometry data

Spirometry is assessed pre-treatment on Week 0, and pre-dose at Weeks 4, 12 and 24.

Spirometry data including FEV1 and FVC will be transferred from the vendor to GSK. When spirometry has been performed but the reading was unacceptable, a record in the database will indicate that the spirometry was performed but all data will be missing and will not be included in listings or summary displays.

The definition of baseline FEV1 and FVC is in Section 10.5.2.1 and of trough FEV1 and FVC is in Section 10.6.4.

## 7.1.2. Planned Efficacy Statistical Analyses

## **Primary Statistical Analyses**

# Endpoint(s)

Trough FEV1

# **Model Specification**

- The primary endpoint of change from baseline in trough FEV1 will be analyzed in the mPP population, using a mixed model repeated measures (MMRM) analysis, including trough FEV1 recorded at each of Week 4, 12 and 24. The model will include covariates of baseline FEV1, stratum (number of long-acting bronchodilators per day during the run-in), Visit, geographical region, treatment and Visit by baseline interaction. A Visit by treatment interaction term will also be included to allow treatment effects to be estimated at each visit separately.
- The variance-covariance matrix will be assumed unstructured.
- Two models will be fitted; one with a response variable of trough FEV1, and one with a response variable of change from baseline in trough FEV1.

# **Handling of Missing Data for Analysis**

 No data were collected for subjects who prematurely discontinued study treatment. All missing and excluded data will be assumed to be Missing at Random (MAR). Sensitivity analyses to investigate the impact of this assumption will be conducted as described below.

# **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Least Square (LS) mean and LS mean change from baseline with their corresponding standard errors (SEs) will be presented for each treatment by Visit, together with estimated treatment differences (FF/UMEC/VI vs. FF/VI+UMEC) and the corresponding 95% confidence intervals (CIs).
- A plot of LS means change from baseline and 95% CIs from the model will be generated for each treatment by Visit.

#### **Example SAS Code**

```
proc mixed data=<dataset>;
    class treatment visit cengroup stratum subjid;
    model endpoint=baseline stratum visit cengroup treatment visit*baseline
    visit*treatment / ddfm=kr;
    repeated visit/ subject=subjid type=un;
    lsmeans visit*treatment / cl diff e om=OMdset at (baseline)=(&blm.);
    ods output lsmeans=lsmeans;
    ods output diffs=diffs;
run;
```

where OMdset is a dataset with a row for every subject-visit combination that contains all of the covariates and blm is a macro variable containing the mean baseline for the subjects used in the analysis. This is used to derive the LS means using coefficients which are based on the subjects used in the analysis.

#### **Sensitivity and Supportive Statistical Analyses**

The above will be repeated for the ITT population. LS mean and LS mean change from

### **Sensitivity and Supportive Statistical Analyses**

baseline with their corresponding SEs will be presented for each treatment by Visit, together with estimated treatment differences and the corresponding 95% CIs.

- A "tipping point" sensitivity analysis of trough FEV1 at Week 24 will be conducted for the mPP Population. This will explore the impact of missing data by using differing assumptions regarding the mean treatment effect in subjects who discontinue study treatment or have data excluded from the mPP Population analyses. Mean treatment effects investigated will range from a change from baseline of -150mL to +150mL in increments of 50mL. For each value of the assumed mean change from baseline on FF/UMEC/VI, the full range of values for the assumed mean change from baseline for FF/VI+UMEC will be investigated; thus including scenarios where subjects who discontinue FF/UMEC/VI have a lower treatment effect than those who discontinue FF/VI+UMEC and vice versa. The analysis results will be used to explore the conditions under which the conclusion of non-inferiority no longer holds.
  - o For each subject with missing or excluded data at Week 24, a value will be imputed based on a random draw from a normal distribution with mean equal to the corresponding assumed mean change from baseline and standard deviation taken from the observed change from baseline data for the combined treatment arms at the Week 24 visit. Data for subjects with missing baseline values will not be imputed. Analysis of the complete Week 24 dataset will be carried out using an ANCOVA model with covariates of treatment group, stratum (number of long-acting bronchodilators per day during the run-in), geographical region and baseline.
  - The seed will be set using the following SAS code:

```
data seed1;
    number=round(10000*ranuni(0),1);
    output;
run;
proc print;
run;
```

The seeds generated and assigned to each analysis will be documented separately prior to DBF.

A table will be produced displaying the 95% CI for the treatment difference at Week 24 under the above assumptions for the mean changes from baseline for each of the treatment arms.

- Interactions between treatment and other factors will be investigated as follows by adding interaction terms to the specified model:
  - An assessment of whether the effect of treatment on trough FEV1 is modified by number
    of long-acting bronchodilators per day during the run-in, geographic region, or baseline will
    be made by fitting separate repeated measures models, identical to the primary analysis
    models described above but also including additional terms as described below.
  - For the factors of number of long-acting bronchodilators per day during the run-in and

#### **Sensitivity and Supportive Statistical Analyses**

geographical region, the primary analysis model will be used with additional terms for the factor by treatment by Visit interaction. The p-value for the treatment by factor interaction at Week 24 will be obtained using contrast statements. If that p-value is  $\geq$  0.10 the interaction will be considered not significant. If the p-value is < 0.10, further investigation will be performed, for example running the analysis by each stratum or geographic region.

○ For baseline FEV1, the primary analysis model will be used with additional terms for the baseline value by treatment by Visit interaction. The p-value for the treatment by baseline interaction at Week 24 will be obtained using contrast statements. If that p-value is ≥ 0.10 the interaction will be considered not significant. If the p-value is < 0.10, further investigation will be performed, for example running the analysis by dichotomous categories of baseline values (values above and below the median).</p>

# 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Other Efficacy Analyses

# 8.1.1. Overview of Planned Efficacy Analyses

The other efficacy analyses will be based on the ITT population, unless otherwise specified.

Table 4 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Section 10.13, List of Data Displays.

Table 4 Overview of Planned Efficacy Analyses

| | | | A | bsolut | te | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Analy | sis | Summary | | Indiv | ridual | Sta | ts Ana | lysis | Summary | | Indiv | idual |
| | Т | F | L | Τ | F | F | L | T | F | L | T | F | F | L |
| SGRQ | | | | | | | | | | | | | | |
| Baseline SGRQ | | | | Υ | | | Υ | | | | | | | |
| Scores | | | | | | | | | | | | | | |
| SGRQ Domain Scores | | | | Υ | | | Υ | | | | Υ | | | |
| SGRQ Total Score | Υ | | | Υ | | | Υ | Υ | Υ | | Υ | <b>Y</b> <sup>2</sup> | | Υ |
| (MMRM Analysis) | | | | | | | | | | | | | | |
| Proportion of | Υ | | | Υ | | | Υ | | | | | | | |
| Responders according | | | | | | | | | | | | | | |
| to SGRQ Total Score | | | | | | | | | | | | | | |
| Baseline Dyspnea Inde | x (BDI | /Trans | sitio | nal Dys | spnea | Inde | x (TDI) | ) | | | | | | |
| BDI | | | | Υ | | | Υ | | | | | | | |
| TDI | Υ | Υ | | Υ | | | Υ | | | | | | | |
| Proportion of | Υ | | | Υ | | | Υ | | | | | | | |
| Responders according | | | | | | | | | | | | | | |
| to TDI Focal Score | | | | | | | | | | | | | | |
| COPD Exacerbations | | | | | | | | | | | | | | |
| Exacerbation | | | | Y1 | | | Υ | | | | | | | |
| Occurrence and | | | | | | | | | | | | | | |
| Details | | | | | | | | | | | | | | |

| | | | Α | bsolut | e | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | sis | Summary | | Individual | | Stats Analysis | | Summary | | Individual | | |
| | T | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| Time to First On-<br>treatment<br>Moderate/Severe<br>Exacerbation | Y | <b>Y</b> <sup>3</sup> | | Y | | | Y | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - Number and percent reporting COPD exacerbation and summary of details regarding the exacerbation. Repeat for post-treatment exacerbations.
  - empirical distribution function plot
  - 3. Kaplan Meier Plot

# 8.1.1.1. St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C)

The SGRQ-C is completed at Week 0, Week 12, and Week 24. The calculation for the SGRQ-C, including how to handle missing values, is detailed in the SGRQ-C manual (Jones, 2016). The conversion of the SGRQ-C scores to SGRQ scores is as described in the manual and as detailed in Section 10.6.4.

Subjects will be classified as responders/non-responders based on SGRQ total score as described in Section 10.6.4

#### 8.1.1.2. COPD Exacerbations

The definition of moderate and severe exacerbations is provided in Section 10.6.4. The definition of on- and post-treatment exacerbations is provided in Section 10.4.2.

For summary of on-treatment COPD exacerbations, details of the event to be summarized include the number and percent of subjects reporting an exacerbation (any severity, mild, moderate, severe and moderate/severe), number and percent subjects with each number of moderate/severe exacerbations  $(0, 1, \ge 2)$ , outcome, severity, duration, whether treatment with systemic or oral steroids was required, whether treatment with antibiotics was required, whether hospitalization was required, and whether the exacerbation resulted in a visit to the emergency room. Post-treatment exacerbations will be similarly summarized. The total number of exacerbations will be included. For derivation of time to first on treatment moderate or severe exacerbation, see Section 10.6.4.

# 8.1.1.3. Baseline Dyspnea Index (BDI)/Transitional Dyspnea Index (TDI) Focal Score

BDI is assessed at Week 0. TDI is assessed at Week 12 and Week 24. The BDI and TDI focal scores [Mahler, 2004] will be calculated as shown in Section 10.6.4.

## 8.1.2. Planned Other Efficacy Statistical Analyses

#### 8.1.2.1. SGRQ Total Score

## **Secondary Statistical Analyses**

# Endpoint(s)

SGRQ total score

# Model Specification, Model Checking & Diagnostics, Model Results Presentation

- Same as for trough FEV1, see Section 7.1.2
- Visit includes week 12 and 24.

#### 8.1.2.2. TDI

#### **Secondary Statistical Analyses**

# **Endpoints**

TDI focal score

# Model Specification, Checking, Results Presentation and SAS code

- Same as for trough FEV1, see Section 7.1.2
- BDI will be used in place of baseline.
- Visit includes week 12 and 24.

# 8.1.2.3. Proportion of Responders according to SGRQ Total Score and Responders according to TDI

#### **Endpoints**

- Proportion of Responders according to SGRQ total score
- Proportion of Responders according to TDI

#### Model Specification

- Generalized Linear Mixed Model
- Terms in the model:

Dependent Variable: Response (Yes/No)

Categorical: treatment group, stratum, geographical region, visit

Continuous: Baseline (for SGRQ total score) or BDI

Interaction: baseline\*Visit.treatment\*Visit

Repeated : Visit

- The model will be fit with an unstructured variance-covariance matrix
- One single model to include all visits
  - SGRQ: include Week 12 and 24
  - TDI: include Week 12 and 24

#### **Handling of Missing Data for Analysis**

- Subjects with missing on-treatment data and a subsequent non-missing on-treatment scheduled assessment will not be considered as a responder/non-responder but will be left as missing.
- Subjects that have withdrawn from the study prior to the visit in question will be imputed as

non-responders at all visits post-withdrawal where the assessment was expected to be performed.

• Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Number and percentage of responders and non-responders for each treatment at each Week
- Odds ratio for comparison between FF/UMEC/VI and FF/VI+UMEC with associated 95% CI

# **Example SAS Code**

run;

#### 8.1.2.4. COPD Exacerbations

# **Secondary Statistical Analyses**

*ods output diffs=differs;* 

## **Endpoints**

• Time to first on-treatment moderate/severe COPD exacerbation

#### **Model Specification**

Cox's proportional hazards model

#### Terms in the model:

Dependent variable: time to first on-treatment moderate/severe exacerbation Categorical: treatment group, gender, exacerbation history (0, 1, >=2 moderate/severe exacerbations in the last 12 month at screening), smoking status (screening), stratum and geographical region.

Continuous: % predicted FEV1 at Baseline

 Use the 'exact' method for handling ties. (If the analysis will not run using the 'exact' method, then the 'Efron' method for handling ties will be used instead.)

#### Handling of Missing Data for Analysis

 Subjects who withdrew from the study prior to experiencing a COPD exacerbation will be considered censored at random.

## **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• Hazard ratio for comparison between FF/UMEC/VI and FF/VI+UMEC with associated 95% CI

# **Example SAS Code**

### **Secondary Statistical Analyses**

proc phreg data=<dataset>;

 $model\ timeto1*eventflag(0)=treatment\ fevpred\ stratum\ cengroup\ smokehis\ hxf\ exac\ /\ risklimits\ ties=exact;$ 

run;

#### **Secondary Statistical Analyses**

### **Endpoints**

• Time to first on-treatment moderate/severe COPD exacerbation

# **Model Specification**

 A Kaplan-Meier analysis will also be performed for figure showing Kaplan-Meier survivor functions of the proportion of subjects with a first exacerbation over time for each treatment group separately plotted on the same figure.

# **Example SAS code**

proc lifetest data=destin outsurv=survest; time timeto1\*eventflag(0);

strata treatment;

run;

#### **Model Results Presentation**

- o Probability of having an event, 95% CI and first quartile time to exacerbation (estimate of the time at which 25% of subjects in each treatment group would have had an exacerbation)
- Figure showing Kaplan-Meier survivor functions of the proportion of subjects with a first exacerbation over time for each treatment group separately plotted on the same figure.

# 8.2. Safety Analyses

# 8.2.1. Overview of Planned Analyses

The safety analyses generally will be based on the ITT population.

Table 5 provides an overview of the planned analyses, with the detailed list of data displays being presented in Section 10.13.

Table 5 Overview of Planned Safety Analyses

| | | Abso | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Indiv | ridual | Sum | mary | Individual | |
| | Т | F | F | L | Т | F | F | Г |
| Exposure | | | | | | | | |
| Exposure Data | Υ | | Υ | Υ | | | | |
| Adverse Events (AEs) | | | | | | | | |
| Overview of On- | Υ | | | | | | | |
| Treatment AEs | | | | | | | | |
| On-Treatment AEs | Y <sup>10</sup> | | | | | | | |
| Post-Treatment AEs | Υ | | | | | | | |
| On-Treatment Drug- | Υ | | | | | | | |
| Related AEs | | | | | | | | |
| Pre-Treatment SAEs | Y1,2 | | | | | | | |

| | | Abs | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sum | mary | | vidual | | nmary | | /idual |
| | T | F | F | L | T | F | F | L |
| On-Treatment SAEs | Υ | | | | | | | |
| Post-Treatment SAEs | Υ | | | | | | | |
| On-Treatment Fatal | Υ | | | | | | | |
| SAEs | | | | | | | | |
| On-Treatment Drug- | Υ | | | | | | | |
| Related SAEs | | | | | | | | |
| Pre-Treatment SAEs | <b>Y</b> 1 | | | | | | | |
| Leading to Withdrawal | | | | | | | | |
| from Study | | | | | | | | |
| On-Treatment AEs | Υ | | | | | | | |
| Leading to Withdrawal | | | | | | | | |
| from Study | | | | | | | | |
| On-Treatment AEs of | Υ | | | | | | | |
| Special Interest On-Treatment SAEs of | Υ | | | | | | | |
| | Y | | | | | | | |
| Special Interest Relationship of AE | <b>Y</b> 1 | | | | | | | |
| System Organ Class, | Ι' | | | | | | | |
| Preferred Term and | | | | | | | | |
| Verbatim Text | | | | | | | | |
| On-treatment Common | Υ | | | | | | | |
| Non-Serious AEs (3% | • | | | | | | | |
| or More of Subjects in | | | | | | | | |
| Any Treatment Group) | | | | | | | | |
| 10 Most Frequent On- | Υ | | | | | | | |
| treatment Adverse | | | | | | | | |
| Event in Each | | | | | | | | |
| Treatment Group | | | | | | | | |
| On-treatment | Υ | | | | | | | |
| Adverse Events by | | | | | | | | |
| System Organ Class | | | | | | | | |
| and Maximum | | | | | | | | |
| Intensity | | | | | | | | |
| Subject Numbers for | | | | Υ1 | | | | |
| Individual AEs | | | | | | | | |
| All AEs | | | | <b>Y</b> 1 | | | | |
| Non-Fatal Serious AEs | | | | Υ1 | | | | |
| Fatal AEs | | | | Υ1 | | | | |
| AEs Leading to | | | | Υ | | | | |
| Withdrawal from Study | | | | ļ ,, | | | | |
| Subject Numbers for | | | | Y | | | | |
| On-Treatment AEs of | | | | | | | | |
| Special Interest | | | | Y | | | | |
| Reasons for | | | | ĭ | | | | |
| Considering as a | | | | | | | | |
| Serious Adverse | | | | | | | | |
| Event | | | | | | | | |

| | Absolute | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Indiv | Individual | | Summary | | Individual |
| | Т | F | F | L | Т | F | F | L |
| Pneumonia | • | | 1 | <u> </u> | | | | • |
| On-Treatment | <b>Y</b> 9 | | | Υ3 | | | | |
| Pneumonias Incidence | | | | | | | | |
| Details of on-treatment | <b>Y</b> 9 | | | Υ3 | | | | |
| Pneumonia | | | | | | | | |
| Post-Treatment | <b>Y</b> 9 | | | Υ3 | | | | |
| Pneumonias Incidence | | | | | | | | |
| Details of Post- | <b>Y</b> 9 | | | <b>Y</b> 3 | | | | |
| treatment Pneumonia | | | | | | | | |
| Bone Fractures | | | | | | | | |
| On-Treatment Bone | Y | | | <b>Y</b> 3 | | | | |
| Fractures | | | | | | | | |
| Post-Treatment Bone | Y | | | <b>Y</b> 3 | | | | |
| Fractures | | | | | | | | |
| Radiography (Chest Im | aging inc | luding X-R | Rays and C | T Scan) | | | | |
| On-Treatment Chest | Y | | | Y3 | | | | |
| Imaging | | | | | | | | |
| Post-Treatment Chest | Υ | | | <b>Y</b> 3 | | | | |
| Imaging | | | | | | | | |
| Liver Events | | | | | | | | |
| Medical conditions | | | | Υ | | | | |
| for subjects with liver | | | | | | | | |
| stopping events | | | | | | | | |
| Liver Event Results | | | | Υ | | | | |
| and Time of Event | | | | | | | | |
| Relative to Treatment | | | | | | | | |
| Liver Event Substance | | | | Υ | | | | |
| Use | | | | | | | | |
| Liver Event Information | | | | Υ | | | | |
| for RUCAM Score | | | | | | | | |
| Liver Biopsy Details | | | | Υ | | | | |
| Liver Imaging Details | | | | Υ | | | | |
| On Treatment Laborato | ry Param | eters | | | | l | | |
| Liver Function Tests | | <b>Y</b> 6 | | | | | | |
| Chemistry Values for | | | | Υ | | | | |
| Subjects with at Least | | | | | | | | |
| One Value Outside the | | | | | | | | |
| Normal Range | | | | | | | | |
| Chemistry Data | Y | Y <sup>4</sup> | | | Υ | <b>Y</b> 5 | | |
| Chemistry Data | Y | | | | | | | |
| Outside the Normal | | | | | | | | |
| Range | | | | | | | | |
| Chemistry Changes | Y | | | | | | | |
| from Baseline Relative | | | | | | | | |
| to the Normal Range | | | | | | | | |
| Hematology Values for | | | | Υ | | | | |
| Subjects with at Least | | | | | | | | |
| One Value Outside the | | | | | | | | |

| | Absolute | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | T | F | F | L | T | F | F | L |
| Normal Range | | | | | | | | |
| Hematology Data | Υ | Y <sup>4</sup> | | | Υ | <b>Y</b> 5 | | |
| Hematology Data | Υ | | | | | | | |
| Outside the Normal | | | | | | | | |
| Range | | | | | | | | |
| Hematology Changes | Υ | | | | | | | |
| from Baseline Relative | | | | | | | | |
| to the Normal Range | | | | | | | | |
| On Treatment Vital Sign | | | | | | | | |
| Vital Sign Data (Pulse | Υ | | | Υ | Υ | | | |
| Rate, Sys BP, Dia BP) | | | | | | | | |
| 12-Lead ECGs | | | | | | _ | | |
| ECG Values | Υ | | | <b>Y</b> <sup>7</sup> | Υ | | Y8 | |
| ECG Findings | Υ | | | | | | | |
| ECG Findings Shifts | Υ | | | | | | | |
| from Baseline | | | | | | | | |
| QTcF Categories | Υ | | | | Υ | | | |
| ECG Abnormalities | Υ | | | <b>Y</b> <sup>7</sup> | | | Y8 | |
| ECG Abnormalities | Υ | | | | | | | |
| Occurring in at least | | | | | | | | |
| 3% of Subjects in | | | | | | | | |
| Either Treatment | | | | | | | | |
| Group | | | | | | | | |
| Maximum Post- | | Υ8 | | | | Y8 | | |
| Baseline QTcF | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. ASE Population
- 2. ITT Population
- 3. Combined listing for on-treatment and post-treatment.
- 4. Separate box plots of change from baseline in maximum and minimum post-baseline values
- 5. Separate scatter plots for maximum and minimum post-baseline versus baseline divided by ULN for maximum and LLN for minimum
- 6. Trellis Display of Maximum Post-baseline Liver Function Test Values Versus Baseline Liver Function Test Values
- 7. Listing of data only for subjects with any abnormal ECG finding.
- 8. Empirical Distribution Function Plot
- 9. Pneumonia are the cases recorded in Pneumonia Details CRF form
- 10. Repeat for by country
- 11. Trellis plot baseline vs post baseline

#### 8.2.1.1. Adverse Events of Special Interest

Adverse events (AEs) of special interest (AESI) have been defined as AEs which have specified areas of interest for FF, VI, or UMEC or for the COPD population. A list of Standardized Medical Dictionary for Regulatory Affairs (MedDRA) Queries (SMQs) and other groupings for AESI is provided in Section 10.6.3.

#### 8.2.1.2. Pneumonia

Summaries of pneumonia will include data from the Pneumonia Details CRF form.

#### **8.2.1.3.** Vital Signs

Vital signs are collected at Screening (Visit 1) and pre-dose at Week 4, Week 24 or at the Early Withdrawal Visit. Vital signs collected at Early Withdrawal and at the onset of a pneumonia event will be included in 'minimum/maximum post-baseline' (see Section 10.6.3 for the definition) summaries but will not be summarized separately.

#### 8.2.1.4. ECGs

12-Lead ECGs are collected at Screening (Visit 1) and approximately 15-45 min after dosing at Week 24 or at the Early Withdrawal Visit. All ECG data present in the database will be considered valid and will be reported (even if the ECG had a technical error). ECGs collected at Study Treatment Discontinuation will be included in summary of ECG finding where 'worst case post-baseline' summarized but will not be summarized separately.

#### 8.2.1.5. Pregnancy

Any pregnancies reported during the study will be summarized in case narratives. Any pregnancy complication or elective termination of a pregnancy for medical reasons will be recorded as an AE or SAE and included in summaries and listings of AEs/SAEs.

# 9. REFERENCES

Aguis R and Kintz P (2010) Drug and alcohol testing in hair, collection and analysis. European workplace drug testing society, version 1.0, 1-18

Barbosa, J, Faria, J, Carvalho, F, Pedro, M, Queiros, O, Moreira, R and Dinis-Oliveira RJ (2013) Hair as an alternative matrix in bioanalysis. Bioanalysis 5 (8):

GlaxoSmithKline Document Number 2015N261999\_03, 200812, A phase IIIB, 24-week randomised, double-blind study to compare 'closed' triple therapy (FF/UMEC/VI) with 'open' triple therapy (FF/VI + UMEC), in subjects with chronic obstructive pulmonary disease (COPD), 26-JUN-2016

GOLD. Global Initiative for Chronic Obstructive Lung Disease (Updated 2015).http://www.goldcopd.org.

Jones, PW and Forde Y (2016). St. Georges Respiratory Questionnaire for COPD Patients Manual, version 1.3.

Mahler DA, Ward J, Fierro-Carrion G, Waterman LA, Lentine TF, Mejia-Alfaro R, Baird JC (2004). Development of Self-Administered Versions of Modified Baseline and Transition Dyspnea Indexes in COPD. COPD Journal of Chronic Obstructive Pulmonary Disease 1(2), pp. 165-172.

Meguro M, Barley EA, Spencer S et al. Development and validation of an improved COPD-Specific Version of the St. George Respiratory Questionnaire. Chest.2007;132:456-463

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for mPP Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Assessment Windows |
| Section 10.4 | Appendix 4: Treatment States & Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.8 | Appendix 8: Multicentre Studies |
| | Laboratory Values |
| | • ECG |
| | Vital Signs |
| Section 10.9 | Appendix 9: Examination of Covariates and Subgroups |
| Section 10.10 | Appendix 10: Multiple Comparisons and Multiplicity |
| Section 10.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 10.12 | Appendix 12: Abbreviations & Trade Marks |
| Section 10.13 | Appendix 13: List of Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for mPP Population

## 10.1.1. Exclusion of Data from the ITT Analyses

In general, all data recorded for subjects who were randomised (excluding those randomised in error) will be included in ITT analyses. The following will result in exclusion of data from ITT analyses:

Spirometry data are excluded from ITT analyses if the actual time of assessment is after the time of dosing on that day or if albuterol/salbutamol was used within 4h of the assessment on that day.

# 10.1.2. Exclusions from mPP Population

The full list of protocol deviations collected on the eCRF is in the PDMP.

The mPP Population is the primary analysis population, comprising all subjects from ITT population with the exception of:

- Full exclusion: subjects who have a full protocol deviation considered to impact primary endpoint (trough FEV1)
  - Eligibility criteria (those that impacts primary endpoint as listed in PDMP, Appendix 2) not met
  - Treatment non-compliance (overall compliance <80% or >120% over the 24-week treatment period, based on active treatment)
  - Randomisation criteria not met
    - Pneumonia or moderate/severe COPD exacerbation during runin
    - Any change to COPD maintenance medications (including dosage and regimen) during the run-in
    - Antibiotics for respiratory tract infections during the run-in
- Partial exclusion: subjects who have a protocol deviation considered to impact primary endpoint. Trough FEV1 assessments collected after the incidence of the protocol deviation will be excluded from primary analysis.
  - Subject received incorrect container which contains incorrect study treatment.
  - Subjects took prohibited medication during treatment period, as detailed in PDMP Appendix 3 Prohibited Medication.

- Partial exclusion: other events (not a protocol deviation) considered to impact the primary endpoint. Trough FEV1 assessments collected on or after the event start date will be excluded from primary analysis.
  - Subjects had a moderate/severe COPD exacerbation
  - Subjects had pneumonia.
  - Subjects who were unblinded by GCSP due to safety concerns.

Note: Subjects who received incorrect treatment and non-compliance based on active treatment will be identified as important PDs and flagged as PP exclusionary following treatment unblinding. These PDs will be flagged as PP exclusionary in ADaM DV dataset and will be included in summary of exclusion from mPP population table.

# 10.2. Appendix 2: Time & Events

| Protocol Activity | Pre-<br>Screen | Screen | Tre | atmei | nt | | Follow Up | |
|---|---|---|---|---|---|---|---|---|
| | Visit 0<br>Pre-<br>screen | Visit 1<br>Screening | Visit 2<br>Randomisation | | Visit<br>4 | Visit 5 | Early<br>Withdrawal<br>Visit | Safety<br>Follow-<br>up<br>Contact |
| Study Week | | Week -2 | Week 0 | Week<br>4 | Week<br>12 | Week<br>24 | | 1 week<br>Fw-up |
| Window | | -3/+8d | | -<br>4/+2d | -8/+6d | -8/+6d | | -1/+4d |
| Written Informed Consent a | Х | Х | | | | | | |
| Genetic Informed Consent b | Χ | Х | | | | | | |
| Demography <sup>c</sup> | Χ | Χ | | | | | | |
| Medical History, including cardiovascular history | | X | | | | | | |
| COPD and Exacerbation<br>History | | Х | | | | | | |
| Concomitant Medication Assessment | Х | Х | х | χ | Х | Х | Х | Х |
| Inclusion/Exclusion Criteria | | Х | | | | | | |
| Randomisation Criteria | | | Х | | | | | |
| Smoking History | | Х | | | | | | |
| Smoking status | | X | | | | Χ | Х | |
| Smoking Cessation | | | | | | | | |
| Counselling | | Χ | | | | X | Х | |
| Register Visit in IRT/ RAMOS | | Х | х | χ | X | Х | Х | |
| Reversibility Testing e | | Х | | | | | | |
| Spirometry | | | <b>Χ</b> f | Χf | Χf | Χf | | |
| Device training and | | | | | | | | |
| registration | | Χ | Х | | | | | |
| Exacerbation Assessment | | Х | Х | Х | Х | Χ | Х | Х |
| SGRQ-C <sup>9</sup> | | | X | | X | X | | |
| BDI <sup>g</sup> | | | Х | | | | | |
| TDI <sup>g</sup> | | | | | Χ | Χ | | |
| CAT <sup>g</sup> | | Х | | | | | | |
| eDevice close out h | | | Х | | | Х | Х | |
| Physical examination i | | Х | | | | X | X | |
| Adverse Events Assessment | | X | Х | Х | Х | X | Х | Х |
| Vital signs j | | X | | X | | X | X | - |
| ECG | | X | | | | Xk | X <sup>k</sup> | |
| Chest X-ray <sup> </sup> | | X | | | | Λ. | | |
| Pulse oximetry m | | ^ | X | | | | | |
| Blood draw for PK | | | ^ | | <b>X</b> n | Χο | | |
| Blood Draw for Genetics | | | | | Λ | | | |
| research | | | | | | Хр | | |

# CONFIDENTIAL

| Protocol Activity | Pre-<br>Screen | Screen | Tre | Follow Up | | | | |
|---|---|---|---|---|---|---|---|---|
| | Visit 0<br>Pre-<br>screen | Visit 1 | Visit 2<br>Randomisation | Visit<br>3 | Visit<br>4 | Visit 5 | Early<br>Withdrawal<br>Visit | Safety<br>Follow-<br>up<br>Contact |
| Study Week | | Week -2 | Week 0 | Week<br>4 | Week<br>12 | Week<br>24 | | 1 week<br>Fw-up |
| Window | | -3/+8d | | -<br>4/+2d | -8/+6d | -8/+6d | | -1/+4d |
| Haematology/biochemistry q | | Х | | | | Χ | Х | |
| Urine Pregnancy Test r | | Х | | Χ | Χ | Х | Χ | |
| Hepatitis B and C tests | | Х | | | | | | |
| Dispense study treatment | | | Х | X | X | | | |
| Administer study treatment in clinic s | | | Х | Х | Х | Х | Х | |
| Assess study treatment compliance | | | | χ | Х | Х | Х | |
| Collect study treatment | | | | Χ | Χ | Χ | Χ | |
| Dispense albuterol/salbutamol | | Х | Х | χ | Х | | | |
| Collect albuterol/salbutamol | | | Х | Χ | Χ | Χ | Χ | |
| Issue/review paper diary t | | Χ | Х | Χ | Χ | Х | Χ | |

- a. Informed consent must be conducted at the Pre-screen Visit prior to performing any study procedures including the changing or withholding of medications. The (IC) may be given at Screening Visit 1 if the subject does not take or has not taken any protocol excluded medications.
- b. Genetics research consent may be obtained at the same time as the study IC and must be obtained prior to obtaining a genetic blood sample.
- Demography may be captured at either the Pre-screen Visit or Screening Visit (for subjects who do not have a Pre-screen Visit).
- d. The IRT will be used for randomisation, emergency unblinding and study treatment supply management (Please refer RAMOS NG IRT manual for more information)
- e. At Screening Visit 1 both pre and post-bronchodilator spirometry will be conducted. Pre-bronchodilator spirometry will be performed prior to the subject taking their morning dose of their usual COPD treatment, between 6am and 11am and after withholding rescue albuterol/salbutamol for ≥4 hours.
- f. At Visits 2-5 (and the Early Withdrawal Visit), pre-bronchodilator spirometry will be performed prior to taking the morning dose of study treatment, between 6am and 11am and after withholding rescue albuterol/salbutamol for ≥4 hours.
- g. Patient reported assessments should be conducted in the following order and before other study assessments: SGRQ-C, BDI/TDI.
- h. Close out eDevice for any subject who fails to randomize, withdraws early, or completes Visit 5.
- i. Physical examination may include height, weight, blood pressure, temperature, heart rate.
- j. Vital signs must be performed prior to spirometry and prior to taking morning dose of study mediation.
- k. ECG to be obtained 15 45 minutes post-dose at treatment Visit 5 and Early Withdrawal Visit (if possible). If a subject is not dosed at Early Withdrawal, then an ECG can be taken at any time during the visit
- I. Chest X-ray (PA and lateral) is required at Screening (or historical x-ray obtained within 3 months prior to Screening) and at anytime there is a suspected pneumonia or a mod/severe exacerbation.
- m. Pulse oximetry must be performed at V2 and anytime there is a suspected pneumonia or a moderate or severe exacerbation.
- PK subset A: PK samples of 120 subjects at selected sites, to be obtained at two time points at Visit 4: pre-dose and in the window 5 to 15 minutes post-dose.
   PK subset B: PK samples of 60 subjects at selected sites, to be obtained and Visit 4: pre-dose, 5-15min, 45-
  - 90min, 2.5-4h, 6-8h, 10-12h, 23-24h post-dose.
- o. PK subset A: PK samples of 120 subjects at selected sites, to be obtained at two time points at Visit 5: 5 to 15 minutes post–dose and 45 to 90 minutes post–dose.
- p. The genetics blood sample should be taken at V5 or at any visit after Randomisation (V2).
- q. Haematology and chemistry panels will include liver chemistry, and potassium and glucose levels.
- r. All female subjects of child bearing potential will have a urine pregnancy test at each visit except Visits 2 and follow-up.
- s. Subjects must withhold their morning dose of study treatment at each clinic visit and not take their study treatment dose until instructed to do so by study staff.
- t. Subjects will be issued a paper diary, at screening and other clinic visits (if required) in order to note any changes to concomitant medications and/or incidence of adverse events that may have occurred between clinic visits.
### 10.3. Appendix 3: Assessment Windows

In general, data will be reported according to the nominal time of clinic visits and assessments as specified in the protocol. For example, if a subject recorded values for the Week 4 visit that were actually made on the 21<sup>st</sup> day of treatment, they will be presented as Week 4 values in the summary tables.

Subjects that permanently stop study medication early between scheduled clinic visits should undergo all assessments listed for the Early Withdrawal Visit. Data collected at this visit will be listed and used in summary or analysis tables as part of the 'worst case post baseline' summary/analysis if appropriate.

Subjects that permanently stop study medication early at the time of a scheduled study visit will have data collected in the eCRF as part of the scheduled study visit.

#### 10.4. Appendix 4: Treatment States and Phases

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment. The 'worst case-post baseline' derivation for summaries of data up to Week 24 will consider all scheduled and unscheduled measurements that have been assigned a treatment phase of 'On-treatment'.

#### 10.4.1. Treatment Phase for Concomitant Medication Data

COPD medication combinations taken at screening will include all COPD medications that were taken on the day of the screening visit, excluding medications that stopped on the day of the screening visit. Calculation of stratum, i.e. long-acting bronchodilator usage per day during the run-in (none, one or two long-acting bronchodilators per day), will also be based on the COPD medication taken on the day of the screening visit. If the calculated stratum is different to the randomized stratum, the calculated stratum will be used as a covariate in all analyses, but both values will be listed. Treatment phases for summaries of COPD and non-COPD concomitant medications will be defined as follows:

| | Treatment Phase | | |
|---|---|---|---|
| Definition | Run-in | On-<br>treatment | Post-<br>treatment |
| Subject did not take study treatment (e.g, run-in failures) and conmed stop date > date of Screening or variable that asks if conmed is ongoing (refer hereafter as goingmed) is "yes" | Y | | |
| (Conmed start date <treatment date="" or<br="" start="">variable that asks if medication taken prior to<br/>study is "yes"(refer hereafter as priormed)) and<br/>date of Screening &lt; conmed stop date<br/><treatment date<="" start="" td=""><td>Y</td><td></td><td></td></treatment></treatment> | Y | | |
| (Conmed start date <treatment and="" date="" date<="" date≤conmed="" date≤treatment="" is="" or="" priormed="" start="" stop="" td="" treatment="" yes)=""><td>Y</td><td>Y</td><td></td></treatment> | Y | Y | |
| (Conmed start date <treatment (conmed="" and="" date="" is="" or="" priormed="" start="" stop="" yes)="">treatment stop date or goingmed is "yes")</treatment> | Υ | Y | Υ |
| (Treatment start date≤conmed start date <treatment (treatment="" and="" date="conmed" date)="" date)<="" date≤conmed="" date≤treatment="" or="" start="" stop="" td="" treatment=""><td></td><td>Y</td><td></td></treatment> | | Y | |
| ([Treatment start date≤conmed start date <treatment [treatment="" and(conmed="" date="" date]="" date])="" or="" start="" stop="">treatment stop date or</treatment> | | Y | Y |

| | Treatment Phase | | |
|---|---|---|---|
| Definition | Run-in | On-<br>treatment | Post-<br>treatment |
| goingmed is Yes) | | | |
| Conmed start≥treatment stop date and treatment start date ≠ treatment stop date | | | Y |

#### NOTES:

- A concomitant medication will be classed in every period of the study in which it was taken (e.g., run-in, ontreatment or post-treatment).
- See Section 10.7.2.1 for handling of partial dates.
- If the study treatment stop date is missing, it will be imputed as described in Section 10.6.1.
- Medications that stopped prior to Screening will not be assigned a treatment phase and will not be summarized.

#### 10.4.2. Treatment Phase for Other Data

Treatment phases for assessments scheduled at a set time will be defined according to the planned relative time of the assessment.

Any events/assessments for subjects not in the ITT population will be assigned a Pretreatment phase.

For all events and assessments where time is recorded, pre-treatment and on-treatment and post-treatment phases will be defined as below:

| Treatment Phase | Definition |
|---|---|
| Pre-treatment | Event onset date/time or assessment date/time < treatment start date/time. |
| On-treatment | Treatment start date/time ≤ event onset date/time or assessment date/time ≤ treatment stop date + 1 day, or any event/assessment with a missing or partial onset date unless there is evidence it was not on-treatment. |
| Post-treatment | Event onset date/time or assessment date/time ≥treatment stop date + 2 and event onset date/time or assessment date/time ≤ study conclusion date Note: the study conclusion date reflects the safety F/U contact for study |
| | treatment completers. |

For all events and assessments (with the exception of concomitant medications) where time is not recorded, the pre-treatment, on-treatment and post-treatment phases will be defined as below:

#### CONFIDENTIAL

| Treatment Phase | Definition |
|---|---|
| Pre-treatment | Event onset date or assessment date < treatment start date. |
| On-treatment | Treatment start date ≤ event onset date or assessment date ≤ treatment stop date + 1 day or any event/assessment with a missing or partial onset date unless there is evidence it was not on-treatment. |
| Post-treatment | Event onset date or assessment date ≥treatment stop date + 2 and event onset date or assessment date ≤ study conclusion date |
| | Note: the study conclusion date reflects the safety F/U contact for study treatment completers. |

## 10.5. Appendix 5: Data Display Standards & Handling Conventions

#### 10.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order [1] |
| 1 | FF/UMEC/VI<br>100mcg/62.5mcg/25mcg + Placebo | FF/UMEC/VI 100/62.5/25 | 1 |
| 2 | FF/VI 100mcg/25mcg + UMEC 62.5mcg | FF/VI 100/25 + UMEC 62.5 | 2 |

#### NOTES:

#### 10.5.2. Baseline Definition & Derivations

#### 10.5.2.1. Baseline Definitions

| Parameter | Study Assessments Collected prior to dosing | | Baseline |
|---|---|---|---|
| | Screening | Week 0 (Pre-Dose) | Definition |
| Efficacy | | | |
| Trough FEV1,<br>Trough FVC | Х | X | Week 0 pre-dose. |
| SGRQ total and domain scores | | Х | Week 0 pre-dose |
| Safety | | | |
| Vitals, Labs, ECGs | X | | Most recent individual value prior to first dose (generally Screening but could be a test repeat). |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

#### 10.5.3. **Reporting Process & Standards**

| Reporting Process | |
|---|---|
| Software | |
| The currently su | The currently supported versions of SAS and TCSG software will be used. |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Area | : /arenv/arprod/gsk2834425/mid200812/final |
| QC Spreadsheet | : /arenv/arwork/gsk2834425/mid200812/documents |
| Analysis Datasets | |

- Analysis datasets will be created according to CDISC standards (SDTM Implementation Guide Version 3.1.3 or higher & AdaM Implementation Guide Version 1.0 or higher).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for the final reporting effort for use in writing the CSR.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the treatment to which the subject was randomized unless otherwise stated. However, there may be additional adhoc displays for individual subjects using the actual treatment received.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places will be adopted for reporting of data based on the raw data collected.
- All data (including data collected post-study treatment discontinuation) will be reported according to the treatment to which the subject was randomized unless otherwise stated. However, there may be additional adhoc displays for individual subjects using the actual treatment received.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places will be adopted for reporting of eCRF data based on the raw data collected.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of decimal places.
- Percentages between 1% and 99%, inclusive, will be rounded to integers. Percentages greater than 0%, but less than 1%, will be reported as <1%, and percentages greater than 99%, but less than 100%, will be reported as >99%. .
- Numeric data will be reported at the precision collected on the eCRF.

#### **Reporting Standards**

• The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of decimal places.

#### **Planned and Actual Time**

- Reporting for tables, figures and statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated. Actual time will be used for calculation of times to events and Kaplan-Meier plots.
- Reporting for listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables except as part of a 'worst case postbaseline' assessment.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

#### 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Study Day**

- Calculated as the number of days from treatment start date :
  - Reference date = missing →
    - → Study Day = missing
  - Reference date < treatment start date → Study Day = reference date treatment start date
  - Reference date ≥ treatment start date → Study Day = reference date treatment start date + 1

#### **Study Treatment Stop Date**

If overall treatment stop date is missing it will be imputed as follows:

- For subjects who attended an Early Withdrawal visit, use the date of the Early Withdrawal visit
- For subjects who attended the last on-treatment visit, use the Visit 5 (Week 24) date
- For subjects who died and did not attend an Early Withdrawal visit or the last on-treatment visit, use the date of death
- For all other subjects, use the last recorded exposure start or stop date

#### **Study and Treatment Completion Definitions**

- A subject is considered to have completed the treatment period if they have not prematurely discontinued IP and attended Visit 5.
- A subject is considered to have completed the study if they either attended Visit 5 or had a phone contact at Visit 5.

#### 10.6.2. Study Population

#### **Demographics**

#### Age

- Age will be calculated based on the Pre-screening visit date
- Birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30JUN'.
- Birth date will be presented in listings as 'YYYY'.

#### Age Category

- Age categories are based on age at Pre-screening and are defined as:
  - ≤64 years
  - 65-74 years,
  - 75-84 years
  - ≥85 years

#### **Demographics**

#### **Body Mass Index**

Calculated as weight (kg) / [height (m)]<sup>2</sup>

#### **Subject Disposition**

#### **Subject Withdrawal**

For Kaplan-Meier plots of subject withdrawal over time, censoring will be performed as follows:
 For subject withdrawal, subjects are represented from their Week 0 date to the date of early withdrawal from the study. Subjects that completed the study are censored at the earliest of the date of completion and day 168.

#### **Smoking Status**

At Screening, subjects who were identified as former smokers but who last smoked within 6 months prior to Screening will be re-classified as current smokers prior to summarizing. Subject listings will include original and re-classified status.

#### Compliance

- ELLIPTA™ inhaler A contains FF/UMEC/VI (for subjects in FF/UMEC/VI treatment group) or FF/VI (for subjects in FF/VI+UMEC treatment group) and has container number with prefix 3.
- ELLIPTA™ inhaler B contains placebo (for subjects in FF/UMEC/VI treatment group) or UMEC (for subjects in FF/VI+UMEC treatment group) and has container number with prefix 4.
- If a dose counter start count is missing then it will be assumed to be 30. If any dose counter stop is missing then the treatment compliance will be set to missing for that subject and for that inhaler.
- Number of doses of study drug taken by each subject from each inhaler = Dose counter startdose counter stop.
- Compliance are calculated as follows:
  - Compliance for Ellipta inhaler A = (dose counter start dose counter stop for inhaler A) x
     100 / (exposure stop date exposure start date +1)
  - Compliance for Ellipta Inhaler B=(dose counter start dose counter stop for Inhaler B) x 100 / (exposure stop date – exposure start date +1)
    - Overall Compliance = (compliance for Inhaler A + compliance for inhaler B with active treatment)/2. That is:
      - For subject in FF/UMEC/VI treatment group, Overall Compliance = compliance for Inhaler A
      - For subject in FF/VI + UMEC treatment group, Overall Compliance = (compliance for Inhaler A + compliance for inhaler B)/2
- Overall compliance and compliance for each inhaler will be categorized as follows:
  - < 80 %
  - $\geq$  80 % to < 95 %
  - $\geq$  95 % to  $\leq$ 105 %
  - >105 % to ≤120 %
  - >120 %.
- If a subject received a treatment other than the randomized treatment during the study, the

#### **Subject Disposition**

compliance will still be calculated using data from all containers received and overall exposure start and stop dates.

#### Long-acting Bronchodilator Usage During the Run-in (Randomisation Stratum)

Randomization stratum, long-acting bronchodilator usage during the run-in, will be derived based on the RMC classification and will be grouped into the following 3 categories:

- None
- One long-acting bronchodilator per day
- Two long-acting bronchodilators per day

Long-acting bronchodilator is defined as any COPD medication in Respiratory Medication Class (MRC) under 'Long-acting beta-2 agonist – Group 2' or 'Long-acting beta-2 agonist – Group 3' or 'Long-acting anticholinergic'.

Based on RAMOS NG record, the number of subjects used none long-acting bronchodilator during run-in is very small (ie. <1% of randomized subjects). Therefore, the combined stratum with 2 categories will be used in the statistical analysis, ie, none and one long-acting bronchodilator per day will be combined into one category in analysis.

Ranodmisation stratum is also collected at randomization in RAMOS NG. Both randomization stratum (derived and collected) will be listed.

#### **Medical Conditions and Concomitant Medications**

#### **Cardiovascular Risk Factors**

Subjects with at least one of the following current or past medical conditions at Screening will be classed as having a cardiovascular (CV) risk factor at screening. The number of CV risk factors at Screening  $(0, 1, \text{ or } \ge 2)$  will be derived.

- Angina pectoris
- Coronary artery disease
- Myocardial infarction
- Arrhythmia
- Congestive heart failure
- Hypertension
- Cerebrovascular accident
- Carotid or aorto-femoral vascular disease,
- Diabetes mellitus
- Hypercholesterolemia

#### **COPD Concomitant medications**

COPD concomitant medications will be grouped into the following RMCs based on pre-defined code lists derived from ATC classifications:

- Antiinfectives (antibiotics, antifungals, antivirals, antiseptics)
- Short-acting anticholinergic

#### **Medical Conditions and Concomitant Medications**

- Short-acting beta-2 agonist
- Long-acting anticholinergic
- Long-acting beta-2 agonist
- Xanthine
- PDE4 Inhibitor
- Corticosteroid inhaled
- Corticosteroid depot
- Corticosteroid systemic oral parenteral and intra-articular
- Corticosteroid other
- Leukotriene receptor antagonist
- Nedocromil or cromolyn sodium
- Mucolytic
- Oxygen
- Other medication given for exacerbation
- Other COPD medication

#### **COPD** medication combination

COPD medications taken on the day of the Screening visit will be grouped into the following categories based on the RMC classification:

- ICS
- LABA
- LAMA
- Xanthine
- PDE4 Inhibitors
- Any combination of the above
- Other
- None

#### **Medical Conditions and Concomitant Medications**

#### **COPD Exacerbation History**

- Individual exacerbations during the 12 months prior to Screening and during the study were to be collected on the eCRF by the Investigator.
- COPD exacerbations with onset date on or after the date of Screening will not be included in
  the counts of number of exacerbations in the past year; all other exacerbations recorded on the
  eCRF will be included in the counts, even if onset/resolution dates are missing or earlier than
  the start of the exact 12 month period prior to Screening.
- COPD exacerbations reported in the past 12 months will be categorized as 0, 1, 2, ≥3
- Number of COPD exacerbations reported in the past 12 months prior to Screening will be summarized according to three categories: moderate COPD exacerbations, severe COPD exacerbations and moderate/severe COPD exacerbations.
  - Moderate COPD exacerbations are defined as exacerbations that required treatment with systemic/oral corticosteroids and/or antibiotics (not involving hospitalization).
  - Severe COPD exacerbations are defined as exacerbations that required in-patient hospitalization.
- Total number of moderate/severe COPD exacerbations are defined as total numbers of moderate and severe COPD exacerbations for each subject.
- Summaries of moderate/severe exacerbations by treatment course are defined as
  exacerbations treated with systemic/oral corticosteroids (with or without antibiotics), and
  exacerbations treated with antibiotics (with or without systemic/oral corticosteroids).

#### **Medical Conditions and Concomitant Medications**

#### COPD Assessment Test (CAT) at Screening

#### **CAT Score**

The CAT consists of eight items each formatted as a six-point differential scale: 0 (no impact) to 5 (high impact). A CAT score will be calculated by summing the non-missing scores on the eight items with a range from 0 to 40. If one item is missing, then the score for that item is set as the average of the non-missing items. If more than one item is missing, then the CAT score will be set to missing.

The CAT score at screening will be summarized.

#### **CAT Category**

Subject will be classified into the following CAT category based on the CAT score at Screening:

- CAT <10</li>
- CAT≥10

The CAT category at screening will be summarised

#### **Baseline Lung Function**

#### Reversibility

The reversibility to salbutamol status of a subject is calculated at Screening and is based on the difference (absolute change and % change) between a subject's pre-salbutamol assessment of FEV1 and their post-salbutamol assessment FEV1 and is defined as follows:

- Reversible, if they had a difference in FEV1 of ≥ 12% and ≥ 200 mL, or
- Non-reversible, if they had a difference in FEV1 of < 200 mL or a ≥ 200 mL difference that was < 12 % of the pre-salbutamol FEV1.</li>

#### **GOLD Grade 1-4 at Screening**

Subjects will be classified into Global Initiative on Obstructive Lung Disease (GOLD) Grades 1-4 using the post-salbutamol percent predicted FEV1 assessment at Screening:

- GOLD Grade 1 (Mild): percent predicted FEV1 ≥ 80%
- GOLD Grade 2 (Moderate): 50%≤ percent predicted FEV1 < 80%</li>
- GOLD Grade 3 (Severe): 30%≤ percent predicted FEV1 < 50%</li>
- GOLD Grade 4 (Very Severe): percent predicted FEV1 < 30%</li>

#### 10.6.3. Safety

#### **Exposure**

#### **Exposure Duration**

Duration of exposure to study treatment is calculated as:

treatment stop date – treatment start date +1.

| <b>Exposure</b> |
|-----------------|
|-----------------|

#### **Exposure Duration**

#### **Exposure Categories**

For the ITT population, the following exposure categories will be derived:
 ≥1 day, ≥4 weeks, ≥8 weeks, ≥12 weeks, ≥16 weeks, ≥20 weeks and ≥24 weeks

#### **Adverse Events**

#### **AEs of Special Interest**

AESI have been defined as AEs which have specified areas of interest for FF, VI or UMEC or
the overall COPD population. The following table presents the AESI groups. Groups which are
not SMQs are made up of a selection of preferred terms (PTs) defined by GSK. The complete
list, including the PTs which contribute to each of the groups will be provided by Global Clinical
Safety and Pharmacovigilance (GCSP) using the MedDRA version current at the time of
reporting. This will be finalized prior to unblinding.

| AE of special interest group | AE special interest subgroup | Sub-SMQ |
|---|---|---|
| Adrenal suppression | | |
| Anticholinergic syndrome (SMQ) | | |
| Asthma/bronchospasm (SMQ) | | |
| Cardiovascular effects | Cardiac arrhythmia | Arrhythmia related investigations, signs and symptoms (SMQ) Bradyarrhythmia terms, nonspecific (SMQ) Conduction defects (SMQ) Disorders of sinus node function (SMQ) Cardiac arrhythmia terms, nonspecific (SMQ) |
| | | Supraventricular tachyarrhythmias (SMQ) Tachyarrhythmia terms, nonspecific (SMQ) Ventricular tachyarrhythmias (SMQ) |
| | Cardiac failure (SMQ) | |
| | Ischaemic heart disease (SMQ) | |
| | Hypertension (SMQ) | |
| | Central nervous system haemorrhages and cerebrovascular conditions (SMQ) | |
| Ocular effects | Glaucoma (SMQ) Lens Disorder (SMQ) | |
| Decreased bone mineral density and associated fractures | Ecito Disordor (Orrig) | |
| Effects on potassium | | |
| Gastrointestinal obstruction (SMQ) | | |

| Hyperglycaemia/new onset diabetes mellitus (SMQ) |
|--------------------------------------------------|
| Hypersensitivity |
| Local steroid effects |
| Pneumonia |
| LRTI excluding pneumonia |
| Tremor |
| Urinary retention |

#### **Bone Fracture Incidents**

If a subject suffers fractures in multiple locations with the same date of fracture, this is considered to be one fracture incident.

All bone fractures will be reported; and separately by traumatic and non-traumatic bone fractures.

| Maximum/Minimum Post-Baseline and Worst-Case Post-Baseline | |
|---|---|
| Definition | Reporting Details |
| Maximum post-baseline;<br>(QTcF, QTcB, PR interval, ECG<br>heart rate, pulse rate, systolic<br>BP, diastolic BP and laboratory<br>tests.) | Maximum on-treatment value over all timepoints. |
| Minimum post-baseline;<br>(Diastolic BP and laboratory<br>tests that do not have a lower<br>limit = 0.) | Minimum on-treatment value over all timepoints. |
| Worst case post-baseline (ECG findings) | <ul> <li>'Abnormal' if any on-treatment assessment is evaluated as 'Abnormal'</li> <li>'Unable to evaluate' if all on-treatment assessments are 'Unable to evaluate'</li> <li>'Normal' if any on-treatment assessment is evaluated as 'Normal' and there are no on-treatment assessments evaluated as 'Abnormal'</li> </ul> |

#### NOTES:

- The treatment phase definitions specified in Section 10.4.2 will be used and only assessments within the ontreatment period will be considered in assessment of minimum/maximum/worst-case post-baseline.
- Assessment of minimum/maximum/worst-case post-baseline will include data from scheduled, unscheduled and study treatment discontinuation visits (if applicable). Vital signs (heart rate, systolic blood pressure and diastolic blood pressure) collected at an assessment associated with a pneumonia event will also be included in derivation of a 'minimum/maximum post-baseline' assessment.

## **Laboratory Parameters**

- Non-quantifiable laboratory results will be treated as missing in summary displays.
   However, the results will be listed as received (e.g. '<x' or '>x').
- An 'any visit post-baseline' classification will be derived, in which subjects will be counted in the 'low' and 'high' categories if they reported a low or high value at any scheduled or

#### **Laboratory Parameters**

unscheduled on-treatment visit during the treatment phase being summarized (see Section 10.4.1 for the definition of treatment phases).

- Change from baseline values will be classified relative to the normal range as 'to low', 'to normal or no change' or 'to high'. Subjects who do not change categories or move from out-of-range to normal will be classified as 'to normal or no change'.
- An 'any visit post-baseline' change classification will be derived, in which subjects will be counted in the 'to low' and 'to high' categories if they reported a change from a 'normal' baseline to a value below or above the normal range (respectively) at any scheduled or unscheduled on-treatment visit during the treatment phase being summarized (see Section 10.4.1 for the definition of treatment phases). Subjects who did not report a change to a value outside the normal range at any visit after the start of study treatment will be counted in the 'to normal or no change' category.

#### Multiple Measurements for Post-Baseline Visits for Safety

 Subjects having both High and Low values relative to Normal Ranges at post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables.

#### **ECG**

QTcF and QTcF change from baseline results will be reported in categories as below:

| ECG Parameter | Units | Ranges | |
|------------------------|-------|--------|-------|
| | | Lower | Upper |
| Absolute | | | |
| | | 0 | ≤ 450 |
| | | > 450 | ≤ 480 |
| Absolute QTcF Interval | msec | > 480 | ≤ 500 |
| | | > 500 | ≤ 530 |
| | | > 530 | |

| ECG | | | |
|---------------------------|--------|------|------|
| Change from Baseline | | | |
| | msec - | | <-60 |
| | | ≥-60 | <-30 |
| Change from Baseline QTcF | | ≥-30 | <0 |
| | | ≥0 | < 30 |
| | | ≥ 30 | <60 |
| | | ≥ 60 | |

#### Association of Chest Imaging (X-ray or CT scan) with Pneumonia Event

- A chest X-ray is considered associated with pneumonia if it is performed within -7 to +14 days
  of the date of onset of pneumonia or the date of resolution, whichever the latter. Pneumonia is
  considered to be supported by a chest X-ray if there is an associated X-ray which shows the
  presence of infiltrates.
- Details of pneumonia events are collected on the Pneumonia Details eCRF page. As there may
  not be a one-to-one correspondence between these events and pneumonia AESI events, a
  cross-tabulation will be provided for the association of pneumonia AESI events and those
  recorded on the Pneumonia Details eCRF page.

### 10.6.4. Efficacy and Health Outcomes

#### Spirometry

Predicted FEV1, Predicted FVC, Absolute and Percent Reversibility in FEV1, Percent Predicted FEV1, Percent Predicted FVC, and Pre-salbutamol and Post-salbutamol FEV1/FVC Ratio

 These derived items will be delivered in a dataset from the vendor for central spirometry, except for post-salbutamol FEV1/FVC ratio, and no recalculation will be performed. Postsalbutamol FEV1/FVC ratio will be calculated as the ratio of post-salbutamol FEV1 and FVC values.

#### **Trough**

- The trough value for FEV1 and FVC at Weeks 4, 12 and 24 is the value of the pre-dose assessment.
- If the actual time of assessment is after the time of dosing on that day, the value for FEV1 and FVC will not be used.
- Change from baseline in trough FEV1 and FVC will be calculated.

#### St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C)

#### General

- The SGRQ-C contains 14 questions with a total of 40 items grouped into three domains (Symptoms, Activity and Impacts).
- The details for how to score the SGRQ-C are outlined in the SGRQ-C manual (Jones, 2016).
   This includes details on how to handle missing data.
- SGRQ-C domain and total score will be converted to SGRQ scores as described in the manual.
- Changes from baseline in domain and total score will be calculated for the converted scores.
- If the language of the SGRQ-C conducted at a post-treatment visit is different to the language used at Day 1, all SGRQ scores at that visit and all subsequent visits will be set to missing.

#### Responder Status according to SGRQ Total Score

- A subject will be a considered a responder according to SGRQ total score if their on-treatment SGRQ total score has decreased at least 4 units from baseline SGRQ total score.
- A subject will be considered a non-responder if their on-treatment SGRQ total score has decreased by less than 4 units, has not changed, or has increased compared to baseline.
- Missing data will be handled as detailed in Section 10.7.2

#### **COPD Exacerbations**

- Each COPD exacerbation will be categorized based on severity as follows:
  - Mild: no treatment with systemic/oral corticosteroids and/or antibiotics and no hospitalization
  - Moderate: required treatment with systemic/oral corticosteroids and/or antibiotics (not involving hospitalization)
  - Severe: required in-patient hospitalization
- The duration of the exacerbation will be calculated as (exacerbation resolution date or date of death exacerbation onset date + 1).
- The time to the first on-treatment exacerbation will be calculated as (exacerbation onset date of first on-treatment exacerbation date of start of treatment + 1).
- Subjects will be represented from their Week 0 date to the earliest of the event or censoring. For subjects who do not experience the event will be censored at the earliest of the date of their treatment stop date +1 day or the date of death.

#### Association to Chest Imaging (X-ray or CT Scan)

 A chest X-ray or CT scan is considered associated with a moderate/severe exacerbation if it is performed within 0 to +14 days of the exacerbation start date.

#### SAC BDI/TDI

#### General

- The BDI focal score will be calculated as the sum of the ratings recorded for each of the three individual scales (Functional Impairment, Magnitude of Task, Magnitude of Effort). Each of these scales has five possible scores ranging from 0 to 4 (with lower scores indicating more impairment), so the range of the BDI focal score is 0 to 12. If a score is missing for any of the three scales, then the BDI focal score will be set to missing. BDI is assessed at baseline (Week 0).
- The SAC TDI focal score will be calculated as the sum of the ratings recorded for each of the three individual scales (Functional Impairment, Magnitude of Task, Magnitude of Effort). Each of these scales has a possible score ranging from -6 to +6. SAC TDI focal score is calculated as the sum of the three individual scores and then divided by 2 (so the range of the TDI focal score is -9 to +9). If a score is missing for any of the three scales, then the SAC TDI focal score will be set to missing.
- If the language of the SAC TDI conducted at a visit is different to the language for the BDI, all TDI scores at that visit and all subsequent visits will be set to missing

#### Responder Status according to SAC TDI Focal Score

- A subject will be a responder if the on-treatment SAC TDI focal score was at least 1 unit at that visit.
- A subject will be considered a non-responder if their on-treatment SAC TDI focal score was less than 1 unit.
- Missing data will be handled as detailed in Section 10.7.2

# 10.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

### 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>For reporting purposes, subject study completion (<i>i.e.</i> as specified in the protocol) was defined as a subject will be considered to have completed the study when they have completed all phases of the study including screening, run-in, randomization, the randomized treatment phase up to visit 5 and safety follow-up visit. Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |
| Vitals/Lab/ECG | Vitals/Lab/ECG data collected as part of the early withdrawal at a scheduled visit, or at a standalone EW visit will be used in the summary of absolute values and change from baseline as part of the 'minimum post baseline', 'minimum change from baseline', 'maximum post-baseline' and 'maximum change from baseline' for diastolic and 'maximum post-baseline' and 'maximum change from baseline' for pulse rate and systolic blood pressure |

## 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> <li>No imputation will be made for any missing numerical data, except in the sensitivity analysis of the primary endpoint to assess the impact of missing data on study results. Missing data will generally not be considered in the calculation of percentages (i.e., the denominator will not include subjects who have missing data at a given time point).</li> </ul> </li> </ul> |
| Responder | <ul> <li>Subjects with a missing baseline will have responder status as missing.</li> <li>Subjects with missing post-baseline data and a subsequent non-missing assessment will not be considered a responder or non-responder but will be left as missing.</li> <li>Subjects with a baseline but all missing post-baseline data will be considered a non-responder at all time points.</li> </ul> |

### 10.7.2.1. Handling of Missing or Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in subject listing displays.</li> <li>Dates which are completely missing will not be imputed, with the exception of the treatment stop date. Details around imputation of the treatment stop date are provided in Section 10.6.1</li> </ul> |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Adverse<br>Events,<br>Exacerbation,<br>Pneumonia | <ul> <li>Any partial dates will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 0 and the event could possibly have occurred during treatment from the partial information, then the Week 0 date will be assumed to be the start date.</li> <li>The event will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> </ul> |
| | <ul> <li>The recorded partial date will be displayed in listings.</li> </ul> |

#### 10.7.2.2. Handling of Missing Data for Statistical Analysis

A "tipping point" sensitivity analysis of trough FEV1 at Week 24 will be conducted for the mPP Population. This will explore the impact of missing data by using differing assumptions regarding the mean treatment effect in subjects who discontinue study treatment or have data excluded from the mPP Population analyses. Further details are given Section 7.1.2.

### 10.8. Appendix 8: Multicenter Studies

## 10.8.1. Methods for Handling Centers

It is likely that many centers will enroll a very small number of subjects and so rather than adjusting for center in the statistical analyses, a geographical region will be used in analyses where specified. The center group will be created based on geographical region and number of randomized subjects in a country, in order to define groups of roughly similar size. The table below shows (most up to date) the numbers in each reagion and the breakdown by stratum.

| Region | Countries | Number of subjects | Number of subjects |
|---|---|---|---|
| | | in each region | in each strata and each region |
| Europe 1 | Russia, Poland<br>Romania | 398 | 0: 9 |
| | | | 1: 195 |
| | | | >=2: 194 |
| | France, Germany,<br>Italy, Spain | 252 | 0: 15 |
| Europe 2 | Europe 2 | | 1: 75 |
| | | | >=2: 162 |
| Asia | Australia, Japan,<br>S. Korea | 215 | 0: 6 |
| | | | 1: 49 |
| | | | >=2: 160 |
| America | Argentina,<br>Mexico | 194 | 0: 3 |
| | | | 1: 139 |
| | | | >=2: 52 |

## 10.9. Appendix 9: Examination of Covariates, Subgroups & Other Strata

#### 10.9.1. Handling of Covariates, Subgroups & Other Strata

- Randomisation is stratified based on long-acting bronchodilator usage during the run-in (none, one or two long-acting bronchodilators per day). The stratum (with none and one combined into the same category based on derived strata) will be fitted as a covariate in all statistical models.
- Other covariates will be included for specific analyses as detailed in model specifications in Section 7 and Section 8.

## 10.10. Appendix 10: Multiple Comparisons & Multiplicity

## 10.10.1. Handling of Multiple Comparisons & Multiplicity

Treatment comparisons will not be adjusted for multiplicity. No p-values for treatment comparisons will be displayed.

## 10.11. Appendix 11: Model Checking and Diagnostics for Statistical Analyses

#### 10.11.1. Statistical Analysis Assumptions

| Endpoints | Trough FEV1 |
|-----------|------------------|
| | SGRQ total score |
| | TDI focal score |
| Analysis | MMRM |

- The Kenward and Roger method (KR) for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
  - O In the event the model fails to run using the KR method, then the residual method will be used instead.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the
  fitted values (i.e. checking the normality assumption and constant variance assumption of
  the model respectively) to gain confidence that the model assumptions are reasonable.

| Endpoints | Proportion of responders according to SGRQ total score, TDI focal score |
|---|---|
| Analysis | Generalized Linear Model |

- Computation of confidence intervals for the odds ratios is based on the individual Wald tests
- FF/VI+UMEC will be used as the reference level for treatment
- Pearson residuals will be plotted by using PLOTS=PEARSONPANEL option for the model statement in SAS.

| Endpoints | Time to first on-treatment moderate/severe COPD exacerbation |
|-----------|--------------------------------------------------------------|
| | • |
| Analysis | Cox's proportional hazard method |

• The proportional hazards assumption for this method of analysis will be examined by obtaining the Kaplan-Meier estimates of the survival function S(t) over time separately for treatment group. Under the assumption of proportional hazard between the treatment groups, In{-In[S(t)]} for the two groups should be parallel to each other and the distance between them constant. If the curves are approximately parallel, then the proportional hazard assumption is not violated. If these curves cross each other or diverge greatly from the assumption of parallel lines, then the assumption is not met.

## 10.12. Appendix 12: Abbreviations

| ADaM | Analysis Data Model |
|---|---|
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ASE | All Subjects Enrolled |
| ATC | |
| BDI | Anatomical Therapeutic Chemical Classification Baseline Dyspnoea Index |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| | Beats Per Minute |
| Bpm | |
| CDISC | COPD Assessment Test |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Intervals |
| COPD | Chronic Obstructive Pulmonary Disease |
| CRT | Case Report Tabulation |
| CSR | Clinical Study Report |
| CRF | Case Report Form |
| CV | Cardiovascular |
| DBF | Database Freeze |
| DM | Data Management |
| DPI | Dry Powder Inhaler |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| FEV1 | Forced Expiratory Volume in One Second |
| FF | Fluticasone Furoate |
| FVC | Forced Vital Capacity |
| GCSP | Global Clinical Safety and Pharmacovigilance |
| GSK | GlaxoSmithKline |
| GSK573719 | Umeclidinium (UMEC) |
| GW642444 | Vilanterol Trifenatate (VI) |
| GW685698 | Fluticasone Furoate (FF) |
| HRQoL | Health Related Quality of Life |
| IB | Investigator Brochure |
| ICS | Inhaled Corticosteroid |
| IDMC | Independent Data Monitoring Committee |
| ITT | Intent-to-Treat |
| LABA | Long Acting Beta-Agonist |
| LAMA | Long-acting Muscarinic Receptor Antagonists |
| MACE | Major Adverse Cardiac Event |
| mcg | Microgram |
| mL | Milliliter |
| MMRM | Mixed Models Repeated Measures |
| mPP | Modified Per-Protocol |
| PD | Protocol Deviation |
| PDMP | |
| LDML | Protocol Deviation Management Plan |

| QD | Once daily |
|------------|--------------------------------------------------------------|
| | , |
| QTc | QT interval corrected for heart rate |
| QTcB | QT interval corrected for heart rate by Bazett's formula |
| QTcF | QT interval corrected for heart rate by Fridericia's formula |
| RAMOS | Randomization & Medication Ordering System |
| RANDALL-NG | GSK Randomization System – Next Generation |
| RAP | Reporting and Analysis Plan |
| RMC | Respiratory Medication Class |
| SABAs | Short-acting β2-adrenergic receptor agonists |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDL | Source Data Lock |
| SDTM | Study Data Tabulation Model |
| SE | Standard Error |
| SGRQ | St Georges Respiratory Questionnaire |
| SGRQ-C | SGRQ for COPD patients |
| SI | System Independent |
| SMQ | Standardized MedDRA Query |
| SOC | System Organ Class |
| TDI | Transitional Dyspnoea Index |
| TFL | Tables, Figures & Listings |
| TSCG | Tibco Spotfire Clinical Graphics software |
| UMEC | Umeclidinium |
| VI | Vilanterol Trifenatate |

## 10.12.1. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| ELLIPTA |
| CAT and COPD Assessment Test |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |

## 10.13. Appendix 13: List of Data Displays

## 10.13.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables Figures | |
|------------------|----------------|-------------|
| Study Population | 1.1 to 1.41 | 1.1 |
| Efficacy | 2.1 to 2.24 | 2.1 to 2.10 |
| Safety | 3.1 to 3.47 | 3.1 to 3.14 |
| Section | Listings | |
| ICH Listings | 1 to 17 | |
| Other Listings | 17 to 50 | |

#### 10.13.2. Programming Note

Unless otherwise stated all listings will be produced by country, treatment, center, and subject. Present Country as a subheading/by variable in listing. In addition, where applicable, listings will include a flag to indicate if the record is on-treatment or post-treatment and a flag to indicate if the subject is in the mPP population.

## 10.13.3. Study Population Tables

| Study | Population Ta | ables | |
|---|---|---|---|
| No. | Populatio<br>n | Title | Deliverable |
| Subjec | t Disposition | | |
| 1.1. | ASE | Summary of Subject Populations and Reason for Screen/Run-in Failure | SAC |
| 1.2. | ITT | Summary of Attendance at Each Visit | SAC |
| 1.3. | ITT | Summary of Completion and Premature Discontinuation of Study Treatment | SAC |
| 1.4. | ITT | Summary of Study Completion and Withdrawal | SAC |
| 1.5. | ASE | Summary of Number of Subjects Enrolled By Country | SAC |
| 1.6. | ASE | Summary of Age ranges | SAC |
| 1.7. | ITT | Summary of Number of Subjects By Geographical Region, Country and Center | SAC |
| 1.8. | MPP | Summary of Number of Subjects By Geographical Region, Country and Center | SAC |
| 1.9. | ASE | Summary of Inclusion/Exclusion Criteria Deviations For Screen Failures | SAC |
| 1.10. | ITT | Summary of Inclusion/Exclusion Criteria Deviations | SAC |
| 1.11. | ITT | Summary of Important Protocol Deviations | SAC |
| 1.12. | ITT | Summary of Exclusions from Modified Per Protocol Population | SAC |
| Demog | raphy | | |
| 1.13. | ITT | Summary of Demographic Characteristics | SAC |
| 1.14. | MPP | Summary of Demographic Characteristics | SAC |
| 1.15. | ITT | Summary of Demographic Characteristics by Country | SAC |
| 1.16. | ITT | Summary of Race and Racial Combinations | SAC |
| 1.17. | MPP | Summary of Race and Racial Combinations | SAC |
| Medica | I Conditions | | |
| 1.18. | ITT | Summary of Current Medical Conditions | SAC |
| 1.19. | ITT | Summary of Past Medical Conditions | SAC |
| 1.20. | ITT | Summary of Cardiovascular Risk Factors | SAC |
| 1.21. | ITT | Summary of Family History of Cardiovascular Risk Factors | SAC |
| 1.22. | ITT | Summary of Smoking History at Screening | SAC |
| Diseas | e Characteris | stics | |
| 1.23. | ITT | Summary of COPD Exacerbation History at Screening | SAC |
| 1.24. | ITT | Summary of Screening Lung Function | SAC |
| 1.25. | MPP | Summary of Screening Lung Function | SAC |
| 1.26. | ITT | Summary of Screening Lung Function by Country | SAC |
| 1.27. | ITT | Summary of Reversibility and GOLD Grade (1-4) at Screening | SAC |
| 1.28. | MPP | Summary of Reversibility and GOLD Grade (1-4) at Screening | SAC |
| 1.29. | ITT | Summary of CAT Score and CAT Category at Screening | SAC |
| Conco | mitant Medic | | |
| 1.30. | ITT | Summary of Long-acting Bronchodilator Usage during the Run-in (Randomization Strata) | SAC |
| 1.31. | MPP | Summary of Long-acting Bronchodilator Usage during the Run-in (Randomization Strata) | SAC |
| 1.32. | ITT | Summary of COPD Concomitant Medication Combinations Taken at Screening | SAC |

| Study | Study Population Tables | | |
|---|---|---|---|
| No. | Populatio<br>n | Title | Deliverable |
| 1.33. | ITT | Summary of COPD Concomitant Medications Taken in the Run-in, Medications Given for Reasons other than an Exacerbation | SAC |
| 1.34. | ITT | Summary of On-Treatment COPD Concomitant Medications,<br>Medications Given for Reasons other than an Exacerbation | SAC |
| 1.35. | ITT | Summary of Post-Treatment COPD Concomitant Medications,<br>Medications Given for Reasons other than an Exacerbation | SAC |
| 1.36. | ITT | Summary of Concomitant Medications Taken in the Run-in Given for An Exacerbation | SAC |
| 1.37. | ITT | Summary of On-Treatment Concomitant Medications Given for an Exacerbation | SAC |
| 1.38. | ITT | Summary of Post-Treatment Concomitant Medications Given For an Exacerbation | SAC |
| 1.39. | ITT | Summary of On-Treatment Non-COPD Concomitant Medications | SAC |
| 1.40. | ITT | Summary of Post-Treatment Non-COPD Concomitant Medications | SAC |
| Treatm | Treatment Compliance | | |
| 1.41. | ITT | Summary of Treatment Compliance (%) | SAC |

## 10.13.4. Study Population Figures

| Study | Study Population figures | | |
|---|---|---|---|
| No. | Populatio<br>n | Title | Deliverable |
| 1.1. | ITT | Kaplan-Meier Plot of Time to Study Withdrawal | SAC |

## 10.13.5. Efficacy Tables

| Efficacy: Tables | | | |
|---|---|---|---|
| No. | Populatio<br>n | Title | Deliverable |
| Spirom | etry | | |
| 2.1 | ITT | Summary of Baseline FEV1 (L) | SAC |
| 2.2 | MPP | Summary of Baseline FEV1 (L) | SAC |
| 2.3. | ITT | Summary of Baseline FEV1 (L) by Country | SAC |
| 2.4. | ITT | Summary of Trough FEV1 (L) | SAC |
| 2.5. | MPP | Summary of Trough FEV1 (L) | SAC |
| 2.6. | ITT | Summary of Trough FEV1 (L) by Country | SAC |
| 2.7. | ITT | Analysis of Trough FEV1 (L) | SAC |
| 2.8. | MPP | Analysis of Trough FEV1 (L) | SAC |
| 2.9. | ITT | Significance Levels for Interactions of Treatment with Number of Long-acting Bronchodilators per Day During the Run-in, Geographical Region, and Baseline for Analysis of Trough FEV1 (L) | SAC |
| 2.10. | mPP | Significance Levels for Interactions of Treatment with Number of Long-acting Bronchodilators per Day During the Run-in, Geographical Region, and Baseline for Analysis of Trough FEV1 (L) | SAC |

| Efficacy | Efficacy: Tables | | |
|---|---|---|---|
| No. | Populatio<br>n | Title | Deliverable |
| 2.11. | MPP | Trough FEV1 (L) Tipping Point Sensitivity Analysis: 95%Cls after Imputing Varying Week 24 Mean Change from Baseline Trough FEV1 (L) | SAC |
| 2.12. | ITT | Summary of Baseline FVC (L) | SAC |
| 2.13. | ITT | Summary of Trough FVC (L) | SAC |
| SGRQ | | | |
| 2.14. | ITT | Summary of Baseline SGRQ Scores | SAC |
| 2.15. | ITT | Summary of SGRQ Scores | SAC |
| 2.16. | ITT | Analysis of SGRQ Total Score | SAC |
| 2.17. | ITT | Summary and Analysis of Proportion of Responders According to SGRQ Total Score | SAC |
| COPD E | xacerbation | S | |
| 2.18. | ITT | Summary of On-Treatment COPD Exacerbations | SAC |
| 2.19. | ITT | Summary of Post-Treatment COPD Exacerbations | SAC |
| 2.20. | ITT | Summary and Analysis of Time to First On-treatment Moderate or Severe Exacerbation (days) | SAC |
| SACBD | I/TDI | | |
| 2.21. | ITT | Summary of SAC BDI Focal Score | SAC |
| 2.22. | ITT | Summary of SAC TDI Focal Score | SAC |
| 2.23. | ITT | Analysis of SAC TDI Focal Score | SAC |
| 2.24. | ITT | Summary and Analysis of Proportion of Responders According to SAC TDI Focal Score | SAC |

## 10.13.6. Efficacy Figures

| Efficad | Efficacy: Figures | | |
|---|---|---|---|
| No. | Populatio<br>n | Title | Deliverable |
| Spiron | netry | | |
| 2.1 | ITT | Box Plot of Change from Baseline in Trough FEV1 (L) at Week 24 | SAC |
| 2.2 | MPP | Box Plot of Change from Baseline in Trough FEV1 (L) at Week 24 | SAC |
| 2.3 | ITT | Empirical Distribution Function Plot of Change from Baseline in Trough FEV1 (L) at Week 24 | SAC |
| 2.4 | MPP | Empirical Distribution Function Plot of Change from Baseline in Trough FEV1 (L) at Week 24 | SAC |
| 2.5 | ITT | Least Squares Mean (95% CI) Change from Baseline in Trough FEV1 (L) | SAC |
| 2.6 | MPP | Least Squares Mean (95% CI) Change from Baseline in Trough FEV1 (L) | SAC |
| SGRQ | | | |
| 2.7 | ITT | Least Squares Mean (95% CI) Change from Baseline in SGRQ Total Score | SAC |
| 2.8 | ITT | Empirical Distribution Function Plot of Change from Baseline in SGRQ Total Score at Week 24 | SAC |
| COPD | COPD Exacerbations | | |
| 2.9 | ITT | Kaplan-Meier Plot of Time to First Moderate/Severe COPD Exacerbation (Days) | SAC |

| Efficac | Efficacy: Figures | | |
|---|---|---|---|
| No. | Populatio<br>n | Title | Deliverable |
| BDI/TD | BDI/TDI | | |
| 2.10 | ITT | Least Squares Means (95% CI) TDI Focal Score | SAC |

## 10.13.7. Safety Tables

| Safety | Safety Tables | | |
|---|---|---|---|
| No. | Population | Title | Deliverable |
| Expos | ure | | |
| 3.1 | ITT | Summary of Exposure | SAC |
| Adver | se Events | | <b> </b> |
| 3.2 | ITT | Overview of On-Treatment Adverse Events | SAC |
| 3.3 | ITT | Summary of On-Treatment Adverse Events | SAC |
| 3.4 | ITT | Summary of On-Treatment Adverse Events by Country | SAC |
| 3.5 | ITT | Summary of Post -Treatment Adverse Events | SAC |
| 3.6 | ITT | Summary of On-treatment Drug-Related Adverse Events | SAC |
| 3.7 | ITT | Summary of Serious Adverse Events (Serious, Drug-Related Serious, Fatal and Drug-Related Serious) by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | SAC |
| 3.8 | ITT | Summary of On-treatment Serious Adverse Events | SAC |
| 3.9 | ITT | Summary of On-treatment Fatal Serious Adverse Events | SAC |
| 3.10 | ASE | Summary of Pre-treatment Serious Adverse Events | SAC |
| 3.11 | ITT | Summary of Pre-treatment Serious Adverse Events | SAC |
| 3.12 | ASE | Summary of Pre-treatment Serious Adverse Events Leading to Withdrawal from Study | SAC |
| 3.13 | ITT | Summary of On-treatment Drug-Related Serious Adverse Events | SAC |
| 3.14 | ITT | Summary of On-treatment Drug-Related Fatal Serious Adverse Events | SAC |
| 3.15 | ITT | Summary of On-treatment Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | SAC |
| 3.16 | ITT | Summary of On-treatment Adverse Events of Special Interest | SAC |
| 3.17 | ITT | Summary of On-treatment Serious Adverse Events of Special Interest | SAC |
| 3.18 | ASE | Relationship of Adverse Event System Organ Class, Preferred Term and Verbatim Text | SAC |
| 3.19 | ITT | Summary of On-Treatment Common (>=3% in Either Treatment Group) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | SAC |
| 3.20 | ITT | Summary of the 10 Most Frequent On-treatment Adverse events in each Treatment Group | SAC |

| Safety | Tables | | |
|---|---|---|---|
| No. | Population | Title | Deliverable |
| 3.21 | ITT | Summary of On-Treatment Adverse Events by System Organ Class and Maximum Intensity | SAC |
| Pneum | ionia | | |
| 3.22 | ITT | Summary of On-treatment Pneumonias Incidence | SAC |
| 3.23 | ITT | Summary of On-treatment Details of Pneumonia | SAC |
| 3.24 | ITT | Summary of Post-treatment Pneumonias | SAC |
| 3.25 | ITT | Summary of Post-treatment Details of Pneumonia | SAC |
| Bone F | ractures | | |
| 3.26 | ITT | Summary of On-treatment Bone Fractures | SAC |
| 3.27 | ITT | Summary of Post-treatment Bone Fractures | SAC |
| Radiog | raphy (Chest | Imaging : X-Rays or CT Scan) | |
| 3.28 | ITT | Summary of On-treatment Chest Imaging (X-Ray or CT Scan | SAC |
| 3.29 | ITT | Summary of Post-treatment Chest Imaging (X-Ray or CT Scan) | SAC |
| Labora | tory Paramete | ers | |
| 3.30 | ITT | Summary of Chemistry Data | SAC |
| 3.31 | ITT | Summary of Change from Baseline in Chemistry Data | SAC |
| 3.32 | ITT | Summary of Chemistry Data Outside the Normal Range | SAC |
| 3.33 | ITT | Summary of Chemistry Changes from Baseline Relative to the Normal Range | SAC |
| 3.34 | ITT | Summary of Hematology Data | SAC |
| 3.35 | ITT | Summary of Change from Baseline in Hematology Data | SAC |
| 3.36 | ITT | Summary of Hematology Data Outside the Normal Range | SAC |
| 3.37 | ITT | Summary of Hematology Changes from Baseline Relative to the Normal Range | SAC |
| Vitals S | Signs | | |
| 3.38 | ITT | Summary of Vital Signs | SAC |
| 3.39 | ITT | Summary of Change from Baseline Vital Signs | SAC |
| ECGs | | | |
| 3.40 | ITT | Summary of ECG Values | SAC |
| 3.41 | ITT | Summary of Change from Baseline in ECG Values | SAC |
| 3.42 | ITT | Summary of QTc(F) (msec) Categories | SAC |
| 3.43 | ITT | Summary of Change From Baseline in QTc(F) (msec) Categories | SAC |
| 3.44 | ITT | Summary of ECG Findings | SAC |
| 3.45 | ITT | Summary of ECG Findings Shifts from Baseline | SAC |
| 3.46 | ITT | Summary of ECG Abnormalities | SAC |

| Safety | Safety Tables | | |
|---|---|---|---|
| No. | Population | Title | Deliverable |
| 3.47 | ITT | Summary of ECG Abnormalities Occurring in at Least 3% of Subjects in Either Treatment Group | SAC |

## 10.13.8. Safety Figures

| Safety | Safety : Figures | | |
|---|---|---|---|
| No. | Popula tion | Title | Deliverable |
| Expos | ure | | |
| 3.1 | ITT | Plot of Exposure to Study Drug | SAC |
| Labora | atory Para | meters | |
| 3.4 | ITT | Trellis Display of Maximum Post-baseline Liver Function Test Values, Versus Baseline Liver Function Test Values | SAC |
| 3.5 | ITT | Scatter Plots of Maximum Post-baseline Versus Baseline For Chemistry Data | SAC |
| 3.6 | ITT | Box Plots of Change from Baseline to Maximum Post-baseline Values for Chemistry Data | SAC |
| 3.7 | ITT | Scatter Plots of Minimum Post-baseline Versus Baseline For Chemistry Data | SAC |
| 3.8 | ITT | Box Plots of Change from Baseline to Minimum Post-baseline Values for Chemistry Data | SAC |
| 3.9 | ITT | Scatter Plots of Maximum Post-baseline Versus Baseline For Hematology Data | SAC |
| 3.10 | ITT | Box Plots of Change from Baseline to Maximum Post-baseline Values for Hematology Data | SAC |
| 3.11 | ITT | Scatter Plots of Minimum Post-baseline Versus Baseline For Hematology Data | SAC |
| 3.12 | ITT | Box Plots of Change from Baseline to Minimum Post-baseline Values for Hematology Data | SAC |
| 12-Lea | d ECGs | | |
| 3.13 | ITT | Empirical Distribution Function Plot of Maximum Post-baseline QTcF (msec) | SAC |
| 3.14 | ITT | Empirical Distribution Function Plot of Change from Baseline in Maximum Post-baseline QTcF (msec) | SAC |

## 10.13.9. ICH Listings

| ICH: | ICH : Listings | | |
|---|---|---|---|
| No. | Popul ation | Title | Deliverable |
| Study | Study population | | |
| 1. | ITT | Listing of Randomized and Actual Treatments | SAC |
| 2. | ITT | Listing of Study Treatment Discontinuation Record | SAC |
| 3. | ITT | Listing of Reasons for Study Withdrawal | SAC |
| 4. | ASE | Listing of Subjects with Inclusion and Exclusion Criteria Deviations for Screen Failures | SAC |
| 5. | ITT | Listing of Subjects with Inclusion and Exclusion Criteria Deviations | SAC |
| 6. | ITT | Listing of Subjects for Whom the Treatment Blind was Broken during the Study | SAC |
| 7. | ITT | Listing of Demographic Characteristics | SAC |
| 8. | ITT | Listing of Race | SAC |
| Spiro | metry | | |
| 9. | ITT | Listing of Raw FEV1 (L) and FVC (L) Data | SAC |
| Expos | sure | | |
| 10. | ITT | Listing of Exposure | SAC |
| Adver | se Event | s | |
| 11. | ASE | Listing of Subject Numbers for Individual Adverse Events | SAC |
| 12. | ASE | Listing of All Adverse Events | SAC |
| 13. | ASE | Listing of Non-Fatal Serious Adverse Events | SAC |
| 14. | ASE | Listing of Fatal Adverse Events | SAC |
| 15. | ITT | Listing of Adverse Events leading to Withdrawal from the Study | SAC |

| ICH : Listings | | | |
|---|---|---|---|
| No. | Popul<br>ation | Title | Deliverable |
| Laboratory Parameters | | | |
| 16. | ITT | Listing of Chemistry Values for Subjects with at Least One Value outside the Normal Range | SAC |
| 17. | ITT | Listing of Hematology Values for Subjects with at Least One Value outside the Normal Range | SAC |

## 10.13.10. Non-ICH Listings

| Non-l | Non-ICH : Listings | | |
|---|---|---|---|
| No. | Popula tion | Title | Deliverable |
| Study | Population | on | |
| 18. | ASE | Listing of Reason for Screen/Run-in Failure | SAC |
| 19. | ITT | Listing of Important Protocol Deviations | SAC |
| 20. | ITT | Listing of Exclusion from Modified Per Protocol Population | SAC |
| 21. | ASE | Listing of Study Treatment Misallocations | SAC |
| 22. | ITT | Listing of Screening Lung Function, Reversibility Status, GOLD Grade and CAT Score | SAC |
| 23. | ITT | Listing of Medical Conditions | SAC |
| 24. | ITT | Listing of Family History of Cardiovascular Risk Factors | SAC |
| 25. | ITT | Listing of COPD Exacerbation History | SAC |
| 26. | ITT | Listing of Smoking History and Smoking Status | SAC |
| 27. | ITT | Listing of Percent Oxygen in Blood | SAC |
| 28. | ITT | Listing of COPD Concomitant Medications | SAC |
| 29. | ITT | Listing of Non-COPD Concomitant Medications | SAC |
| 30. | ITT | Listing of Randomisation Strata (Derived and from eCRF) | SAC |
| 31. | ITT | Relationship between ATC Level 1, Ingredient and Verbatim Text for Non-COPD Medications | SAC |
| 32. | ITT | Listing of Treatment Compliance Data | SAC |

| Non-I | Non-ICH : Listings | | |
|---|---|---|---|
| No. | Popula tion | Title | Deliverable |
| Adver | se Events | | |
| 33. | ITT | Listing of Subject Numbers for On-Treatment Adverse Events of Special Interest | SAC |
| 34. | ITT | Listing of Reasons for Considering as a Serious Adverse Event | SAC |
| COPD | Exacerba | tions | |
| 35. | ITT | Listing of COPD Exacerbations | SAC |
| SGRQ | | | |
| 36. | ITT | Listing of SGRQ Scores | SAC |
| BDI/TI | OI . | | |
| 37. | ITT | Listing of BDI/TDI Focal Scores | SAC |
| CAT | | | |
| 38. | ITT | Listing of CAT Scores | SAC |
| Pneun | nonia Inci | dence | |
| 39. | ITT | Listing of Pneumonia Data | SAC |
| Bone | Fractures | | 1 |
| 40. | ITT | Listing of Bone Fracture Data | SAC |
| Chest | Imaging ( | X-Rays or CT Scan) | 1 |
| 41. | ITT | Listing of Chest Imaging (X-Ray or CT Scan) Data | SAC |
| Liver I | Events | | 1 |
| 42. | ITT | Listing of Liver Event Results and Time of Event Relative to Treatment | SAC |
| 43. | ITT | Listing of Medical Conditions for Subjects with Liver Stopping Events | SAC |
| 44. | ITT | Listing of Substance Use for Subjects with Liver Stopping Events | SAC |
| 45. | ITT | Listing of Liver Event Information for RUCAM Score | SAC |
| 46. | ITT | Listing of Liver Biopsy Details | SAC |
| 47. | ITT | Listing of Liver Imaging Details | SAC |

#### CONFIDENTIAL

| Non-ICH: Listings | | | |
|---|---|---|---|
| No. | Popula<br>tion | Title | Deliverable |
| 12-Lead ECGs | | | |
| 48. | ITT | Listing of ECG Values for Subjects with Any Abnormal ECG Finding | SAC |
| 49. | ITT | Listing of ECG Abnormalities | SAC |
| Inhaler malfunctions | | | |
| 50. | ITT | Listing of Inhaler Malfunctions | SAC |